Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines – Methotrexate vs Hydroxychloroquine

NCT04691505

December 30, 2020

### 1. Comparison Details

#### a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>methotrexate versus</u> <u>hydroxychloroquine</u> for rheumatoid arthritis.

### b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

### 2. Person responsible for implementation of replication in Aetion

Mufaddal Mahesri

### 3. Data Source(s)

Medicare, 2007-2017

### 4. Study Design Diagrams





#### 5. Cohort Identification

#### a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing methotrexate to hydroxychloroquine. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of methotrexate or hydroxychloroquine (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

#### b. Key details regarding cohort creation

#### Index date:

Day of initiation of new methotrexate or hydroxychloroguine use

#### Inclusion criteria for analyses 1, 3, 4:

- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of methotrexate or hydroxychloroquine any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least one inpatient or one outpatient claim with rheumatoid arthritis diagnosis recorded in 365 days prior to and including index date
- No history of nursing home admission recorded in 365 days prior to and including index date
- No use of any DMARDs any time prior to and including index date

#### Inclusion criteria for analysis 2:

- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of tofacitinib or abatacept any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least one inpatient or one outpatient claim with rheumatoid arthritis diagnosis recorded in 365 days prior to and including index date
- 180-day continuous use of tofacitinib or abatacept starting on the index date
- No history of nursing home admission recorded in 365 days prior to and including index date
- No use of any DMARDs any time prior to and including index date

# c. Flowchart of the study cohort assembly

| | Less Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 7,964,044 |
| Did not meet cohort entry criteria | -7,082,612 | 881,432 |
| Excluded due to insufficient enrollment | -334,379 | 547,053 |
| Excluded due to prior use of referent | -157,248 | 389,805 |
| Excluded due to prior use of exposure | -232,714 | 157,091 |
| Excluded because patient qualified in >1 exposure category | -259 | 156,832 |
| Excluded based on Dementia Exclusion | -3,864 | 152,968 |
| Excluded based on RA Diagnosis | -8,284 | 144,684 |
| Excluded based on Nursing Home Admission | -1,513 | 143,171 |
| Excluded based on DMARD use (all DMARDs) | -8,681 | 134,490 |
| Excluded because patient did not begin follow-up | -937 | 133,553 |
| Patients in methotrexate group | | 74,719 |
| Patients in hydroxychloroquine group | | 58,834 |
| Final cohort | | 133,553 |

## 6. Variables

## a. Exposure-related variables:

## Study drug:

The study exposure of interest is initiation of methotrexate

## Comparator:

Initiators of methotrexate will be compared to initiators of hydroxychloroquine

# b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------|------------------|
| Diabetes | Depression |
| Obesity | Anxiety |
| Hypertension | Bipolar disorder |
| Coronary artery disease | Schizophrenia |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking Number of hospitalizations | |
| Mammography | Number of physician office visits |
| Colonoscopy | Number of serum creatinine tests ordered |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination | Number of rheumatologist visits |
| Pneumococcal vaccination | Number of C-reactive protein tests ordered |
| Herpes zoster vaccination | Osteoporosis |

| Bone mineral density test | Fractures |
|-----------------------------------|----------------------------|
| Number of distinct generic agents | Falls |
| Number of emergency room visits | Use of supplemental oxygen |
| Number of outpatient visits | Combined comorbidity score |

| Comedication use | |
|---|---|
| Lithium | Angiotensin II receptor blockers |
| Anti-epileptic mood stabilizers | Angiotensin converting enzyme inhibitors |
| Anti-epileptics (other than mood stabilizers) | Beta blockers |
| Atypical antipsychotics | Calcium channel blockers |
| Benzodiazepines | Diuretics |
| Serotonin-norepinephrine reuptake Inhibitors | Nitrates |
| Selective serotonin reuptake inhibitors | Lipid lowering drugs |
| Tricyclic antidepressants (TCAs) | Non-insulin diabetes medications |
| Typical antipsychotics | Insulin |
| Anticoagulants | Antidepressants |
| Antiplatelet agents | |

| Rheumatoid arthritis related factors | |
|--------------------------------------|---------------------|
| NSAIDs / coxibs | Glucocorticoid dose |
| Opioids | |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Renal dysfunction |
| Coronary artery disease | Chronic liver disease |
| Heart failure | Asthma |
| Stroke or transient ischemic attack | Ischemic heart disease |
| Peripheral vascular disease | Chronic obstructive pulmonary disease |
| Hypertension | Malignancy |
| Diabetes | Drug or alcohol abuse or dependence |
| Hyperlipidemia | Venous thromboembolism |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component:

Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of methotrexate and hydroxychloroquine and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- · End of the study period,
- Measured death event occurs,
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (methotrexate and hydroxychloroquine) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of methotrexate and hydroxychloroquine and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

# 7. Feasibility counts

| Analysis scheme | Total methotrexate /<br>hydroxychloroquine<br>initiators | N outcome | Dementia Rate per 1,000<br>person-years (95% CI) | Follow-up time in days;<br>Median [IQR] |
|---|---|---|---|---|
| 1: As treated | 74,719 (60.5%) | 2,875 | 14.55 (14.02, 15.08) | 227 [02 741] |
| | 58,834 (39.5%) | 2,075 | 14.55 (14.02, 15.06) | 237 [83, 741] |
| 2: 6 mo induction period, 'as started' | 45,480 (58.3%) | 2 212 | 18.87 (18.23, 19.51) | 1,095 [573, 1,095] |
| | 32,530 (41.7%) | 3,313 | 10.07 (10.25, 19.51) | |
| 3: exclude 6 mo follow-up (symptoms to | 44,240 (58.3%) | 2,442 | 16 47 (15 92) | 4E0 [146 1 030] |
| claims period) | 31,645 (41.7%) | 2,442 | 16.47 (15.83) | 458 [146, 1,028] |
| 4: Outcome Dx + Rx | 74,719 (60.5%) | 1 102 | 5.53 (5.20, 5.85) | 220 [02 747] |
| | 58,834 (39.5%) | 1,102 | | 239 [83, 747] |

#### 8. Propensity score analysis

We will use a propensity-score (PS)¹-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.² Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,³ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁴

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>5</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>6</sup>

## a. PS distributions stratified by treatment group

# Pre-matching propensity score overlap:



## Post-matching propensity score overlap:



# b. Table for covariate balance

| | Unmatched | | | | PS-Matched | |
|---|---|---|---|---|---|---|
| Variable | Methotrexate<br>(N = 74,719) | Hydroxychloroquine<br>(N = 58,834) | St. Diff | Methotrexate<br>(N = 54,562) | Hydroxychloroquine<br>(N = 54,562) | St. Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 73.65 (6.39) | 73.79 (6.53) | -0.02 | 73.77 (6.44) | 73.77 (6.53) | 0.00 |
| Gender, n (%) | | | | | | |
| Male | 21,458 (28.7%) | 13,294 (22.6%) | 0.14 | 12,955 (23.7%) | 13,035 (23.9%) | 0.00 |
| Female | 53,261 (71.3%) | 45,540 (77.4%) | -0.14 | 41,607 (76.3%) | 41,527 (76.1%) | 0.00 |
| Race, n (%) | | | | | | |
| White | 62,760 (84.0%) | 49,973 (84.9%) | -0.02 | 46,153 (84.6%) | 46,202 (84.7%) | 0.00 |
| Black | 6,876 (9.2%) | 5,120 (8.7%) | 0.02 | 4,839 (8.9%) | 4,833 (8.9%) | 0.00 |
| Asian | 1,226 (1.6%) | 903 (1.5%) | 0.01 | 861 (1.6%) | 848 (1.6%) | 0.00 |
| Hispanic | 1,923 (2.6%) | 1,402 (2.4%) | 0.01 | 1,372 (2.5%) | 1,335 (2.4%) | 0.01 |
| Native American | 517 (0.7%) | 352 (0.6%) | 0.01 | 329 (0.6%) | 334 (0.6%) | 0.00 |
| Other | 1,039 (1.4%) | 766 (1.3%) | 0.01 | 707 (1.3%) | 718 (1.3%) | 0.00 |
| Unknown | 378 (0.5%) | 318 (0.5%) | 0.00 | 301 (0.6%) | 292 (0.5%) | 0.01 |
| Region, n (%) | | | | | | |
| Northeast | 13,068 (17.5%) | 11,161 (19.0%) | -0.04 | 10,196 (18.7%) | 10,182 (18.7%) | 0.00 |
| South | 32,015 (42.8%) | 25,230 (42.9%) | 0.00 | 23,358 (42.8%) | 23,360 (42.8%) | 0.00 |
| North Central | 16,684 (22.3%) | 12,843 (21.8%) | 0.01 | 11,981 (22.0%) | 12,029 (22.0%) | 0.00 |
| West | 12,700 (17.0%) | 9,484 (16.1%) | 0.02 | 8,912 (16.3%) | 8,876 (16.3%) | 0.00 |
| Unknown | 252 (0.3%) | 116 (0.2%) | 0.02 | 115 (0.2%) | 115 (0.2%) | 0.00 |
| Calendar year of index date, n (%) | | | | | | |
| 2007 | 7,465 (10.0%) | 4,407 (7.5%) | 0.09 | 4,374 (8.0%) | 4,363 (8.0%) | 0.00 |
| 2008 | 3,811 (5.1%) | 2,106 (3.6%) | 0.07 | 2,137 (3.9%) | 2,098 (3.8%) | 0.01 |
| 2009 | 8,055 (10.8%) | 5,824 (9.9%) | 0.03 | 5,525 (10.1%) | 5,573 (10.2%) | 0.00 |

| 2010 | 7,445 (10.0%) | 5,498 (9.3%) | 0.02 | 5,217 (9.6%) | 5,249 (9.6%) | 0.00 |
|---|---|---|---|---|---|---|
| 2011 | 7,570 (10.1%) | 5,741 (9.8%) | 0.01 | 5,431 (10.0%) | 5,433 (10.0%) | 0.00 |
| 2012 | 7,313 (9.8%) | 6,000 (10.2%) | -0.01 | 5,572 (10.2%) | 5,552 (10.2%) | 0.00 |
| 2013 | 7,324 (9.8%) | 6,277 (10.7%) | -0.03 | 5,717 (10.5%) | 5,737 (10.5%) | 0.00 |
| 2014 | 3,573 (4.8%) | 3,330 (5.7%) | -0.04 | 2,959 (5.4%) | 2,939 (5.4%) | 0.00 |
| 2015 | 8,908 (11.9%) | 8,041 (13.7%) | -0.05 | 7,153 (13.1%) | 7,171 (13.1%) | 0.00 |
| 2016 | 3,979 (5.3%) | 3,600 (6.1%) | -0.03 | 3,200 (5.9%) | 3,207 (5.9%) | 0.00 |
| 2017 | 9,276 (12.4%) | 8,010 (13.6%) | -0.04 | 7,277 (13.3%) | 7,240 (13.3%) | 0.00 |
| Low income subsidy, n (%) | 16,327 (21.9%) | 12,143 (20.6%) | 0.03 | 11,388 (20.9%) | 11,430 (20.9%) | 0.00 |
| Dementia risk factors, n (%) | | | | | | |
| Diabetes | 25,372 (34.0%) | 19,427 (33.0%) | 0.02 | 18,092 (33.2%) | 18,047 (33.1%) | 0.00 |
| Obesity | 8,878 (11.9%) | 7,608 (12.9%) | -0.03 | 6,850 (12.6%) | 6,867 (12.6%) | 0.00 |
| Hypertension | 59,412 (79.5%) | 47,473 (80.7%) | -0.03 | 43,928 (80.5%) | 43,816 (80.3%) | 0.01 |
| Coronary artery disease | 20,997 (28.1%) | 16,849 (28.6%) | -0.01 | 15,454 (28.3%) | 15,467 (28.3%) | 0.00 |
| Depression | 11,224 (15.0%) | 10,107 (17.2%) | -0.06 | 8,997 (16.5%) | 8,995 (16.5%) | 0.00 |
| Anxiety | 8,993 (12.0%) | 8,333 (14.2%) | -0.07 | 7,334 (13.4%) | 7,353 (13.5%) | 0.00 |
| Bipolar disorder | 652 (0.9%) | 649 (1.1%) | -0.02 | 552 (1.0%) | 559 (1.0%) | 0.00 |
| Schizophrenia | 213 (0.3%) | 181 (0.3%) | 0.00 | 164 (0.3%) | 162 (0.3%) | 0.00 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Smoking, n (%) | 12,540 (16.8%) | 9,925 (16.9%) | 0.00 | 9,093 (16.7%) | 9,208 (16.9%) | -0.01 |
| Mammography, n (%) | 18,984 (25.4%) | 18,256 (31.0%) | -0.12 | 16,162 (29.6%) | 16,084 (29.5%) | 0.00 |
| Colonoscopy, n (%) | 8,693 (11.6%) | 7,335 (12.5%) | -0.03 | 6,632 (12.2%) | 6,638 (12.2%) | 0.00 |
| Fecal occult blood test, n (%) | 7,166 (9.6%) | 6,189 (10.5%) | -0.03 | 5,556 (10.2%) | 5,578 (10.2%) | 0.00 |
| Influenza vaccination, n (%) | 44,753 (59.9%) | 37,288 (63.4%) | -0.07 | 34,075 (62.5%) | 34,120 (62.5%) | 0.00 |
| Pneumococcal vaccination, n (%) | 14,977 (20.0%) | 13,135 (22.3%) | -0.06 | 11,819 (21.7%) | 11,820 (21.7%) | 0.00 |
| Herpes zoster vaccination, n (%) | 421 (0.6%) | 376 (0.6%) | 0.00 | 349 (0.6%) | 344 (0.6%) | 0.00 |
| Bone mineral density test, n (%) | 17,615 (23.6%) | 14,992 (25.5%) | -0.04 | 13,596 (24.9%) | 13,622 (25.0%) | 0.00 |

| Number of distinct generic agents, | | | | | | |
|---|---|---|---|---|---|---|
| mean (SD) | 12.60 (6.29) | 13.23 (6.39) | 0.00 | 13.03 (6.52) | 13.01 (6.23) | 0.00 |
| Number of emergency room visits, | | | | | | |
| mean (SD) | 0.63 (1.27) | 0.65 (1.31) | 0.00 | 0.64 (1.29) | 0.64 (1.29) | 0.00 |
| Number of outpatient visits, mean | | | | | | |
| (SD) | 16.39 (16.86) | 17.24 (16.62) | 0.00 | 16.90 (17.36) | 16.90 (16.01) | 0.00 |
| Number of hospitalizations, mean | | | | | | |
| (SD) | 0.29 (0.71) | 0.30 (0.74) | 0.00 | 0.30 (0.71) | 0.30 (0.73) | 0.00 |
| Number of physician office visits, | () | | | ( ) | () | |
| mean (SD) | 5.77 (9.76) | 5.72 (9.09) | 0.00 | 5.73 (9.09) | 5.72 (9.19) | 0.00 |
| Number of rheumatologist visits, | 2 22 (2 25) | 2 22 (2 42) | 0.00 | 2 22 (2 24) | 2 22 (2 42) | 0.00 |
| mean (SD) | 2.22 (2.35) | 2.20 (2.10) | 0.00 | 2.20 (2.34) | 2.20 (2.10) | 0.00 |
| Number of C-reactive protein tests | 1 42 /1 66\ | 1 21 /1 44\ | 0.00 | 1 24 (1 52) | 1 24 (1 47) | 0.00 |
| ordered, mean (SD) Number of serum creatinine tests | 1.43 (1.66) | 1.31 (1.44) | 0.00 | 1.34 (1.53) | 1.34 (1.47) | 0.00 |
| ordered, mean (SD) | 3.98 (2.92) | 3.97 (3.09) | 0.00 | 3.97 (2.85) | 3.96 (3.10) | 0.00 |
| Composite frailty score, mean (SD) | 0.16 (0.04) | 0.16 (0.04) | 0.00 | 0.16 (0.04) | 0.16 (0.04) | 0.00 |
| Osteoporosis, n (%) | 21,166 (28.3%) | 17,521 (29.8%) | -0.03 | 16,047 (29.4%) | 16,067 (29.4%) | 0.00 |
| Fractures, n (%) | 6,216 (8.3%) | 5,185 (8.8%) | -0.02 | 4,742 (8.7%) | 4,742 (8.7%) | 0.00 |
| Falls, n (%) | 2,960 (4.0%) | 2,502 (4.3%) | -0.02 | 2,273 (4.2%) | 2,269 (4.2%) | 0.00 |
| Use of supplemental oxygen, n (%) | 686 (0.9%) | 785 (1.3%) | -0.04 | 618 (1.1%) | 648 (1.2%) | -0.01 |
| Combined comorbidity score, mean | (0.075) | 7 00 (2.070) | | 010 (1.179) | 0.0(2.2/3) | 0.02 |
| (SD) | 1.38 (2.20) | 1.60 (2.36) | 0.00 | 1.51 (2.28) | 1.52 (2.30) | 0.00 |
| Comedication use, n (%) | | | | | | |
| Lithium | 93 (0.1%) | 83 (0.1%) | 0.00 | 70 (0.1%) | 72 (0.1%) | 0.00 |
| Anti-epileptic mood stabilizers | 853 (1.1%) | 796 (1.4%) | -0.03 | 688 (1.3%) | 704 (1.3%) | 0.00 |
| Anti-epileptics (other than mood | | | | | | |
| stabilizers) | 13,247 (17.7%) | 12,475 (21.2%) | -0.09 | 10,893 (20.0%) | 10,900 (20.0%) | 0.00 |
| Atypical antipsychotics | 1,088 (1.5%) | 987 (1.7%) | -0.02 | 864 (1.6%) | 875 (1.6%) | 0.00 |
| Benzodiazepines | 6,971 (9.3%) | 6,781 (11.5%) | -0.07 | 5,879 (10.8%) | 5,845 (10.7%) | 0.00 |
| Serotonin-norepinephrine reuptake | . , | | | , | , | |
| inhibitors | 4,980 (6.7%) | 5,150 (8.8%) | -0.08 | 4,330 (7.9%) | 4,353 (8.0%) | 0.00 |

| Selective serotonin reuptake | | | | | | |
|---|---|---|---|---|---|---|
| inhibitors | 12,538 (16.8%) | 10,861 (18.5%) | -0.04 | 9,826 (18.0%) | 9,843 (18.0%) | 0.00 |
| Tricyclic antidepressants (TCAs) | 4,127 (5.5%) | 3,770 (6.4%) | -0.04 | 3,350 (6.1%) | 3,329 (6.1%) | 0.00 |
| Typical antipsychotics | 206 (0.3%) | 147 (0.2%) | 0.02 | 137 (0.3%) | 138 (0.3%) | 0.00 |
| Anticoagulants | 7,753 (10.4%) | 6,473 (11.0%) | -0.02 | 5,912 (10.8%) | 5,903 (10.8%) | 0.00 |
| Antiplatelet agents | 7,013 (9.4%) | 5,346 (9.1%) | 0.01 | 4,989 (9.1%) | 4,964 (9.1%) | 0.00 |
| Angiotensin II receptor blockers | 16,370 (21.9%) | 13,993 (23.8%) | -0.05 | 12,736 (23.3%) | 12,648 (23.2%) | 0.00 |
| Angiotensin converting enzyme | | | | | | |
| inhibitors | 23,816 (31.9%) | 17,848 (30.3%) | 0.03 | 16,882 (30.9%) | 16,802 (30.8%) | 0.00 |
| Beta blockers | 29,260 (39.2%) | 23,690 (40.3%) | -0.02 | 21,943 (40.2%) | 21,770 (39.9%) | 0.01 |
| Calcium channel blockers | 21,542 (28.8%) | 18,133 (30.8%) | -0.04 | 16,525 (30.3%) | 16,530 (30.3%) | 0.00 |
| Diuretics | 23,803 (31.9%) | 19,617 (33.3%) | -0.03 | 17,951 (32.9%) | 17,928 (32.9%) | 0.00 |
| Nitrates | 5,508 (7.4%) | 4,496 (7.6%) | -0.01 | 4,100 (7.5%) | 4,099 (7.5%) | 0.00 |
| Lipid lowering drugs | 37,971 (50.8%) | 30,921 (52.6%) | -0.04 | 28,541 (52.3%) | 28,344 (51.9%) | 0.01 |
| Non-insulin diabetes medications | 14,027 (18.8%) | 10,032 (17.1%) | 0.04 | 9,493 (17.4%) | 9,458 (17.3%) | 0.00 |
| Insulin | 4,493 (6.0%) | 3,579 (6.1%) | 0.00 | 3,334 (6.1%) | 3,264 (6.0%) | 0.00 |
| Antidepressants | 21,471 (28.7%) | 19,536 (33.2%) | -0.10 | 17,319 (31.7%) | 17,308 (31.7%) | 0.00 |
| Rheumatoid arthritis related factors | | | | | | |
| Nonsteroidal anti-inflammatory | | | | | | |
| drugs/Coxibs, n (%) | 33,921 (45.4%) | 25,147 (42.7%) | 0.05 | 23,787 (43.6%) | 23,791 (43.6%) | 0.00 |
| Opioids, n (%) | 48,221 (64.5%) | 37,621 (63.9%) | 0.01 | 34,922 (64.0%) | 34,968 (64.1%) | 0.00 |
| Glucocorticoids use/dose, n (%) | 52,804 (70.7%) | 37,351 (63.5%) | 0.15 | 35,997 (66.0%) | 36,011 (66.0%) | 0.00 |
| Comorbid conditions, n (%) | | | | | | |
| Atrial fibrillation | 8,691 (11.6%) | 7,181 (12.2%) | -0.02 | 6,568 (12.0%) | 6,573 (12.0%) | 0.00 |
| Heart failure | 8,954 (12.0%) | 7,524 (12.8%) | -0.02 | 6,768 (12.4%) | 6,805 (12.5%) | 0.00 |
| Stroke or transient ischemic attack | 6,579 (8.8%) | 5,444 (9.3%) | -0.02 | 4,946 (9.1%) | 4,943 (9.1%) | 0.00 |
| Peripheral vascular disease | 9,374 (12.5%) | 7,837 (13.3%) | -0.02 | 7,131 (13.1%) | 7,142 (13.1%) | 0.00 |
| Hyperlipidemia | 53,606 (71.7%) | 43,255 (73.5%) | -0.04 | 39,871 (73.1%) | 39,833 (73.0%) | 0.00 |

| Renal dysfunction | 9,448 (12.6%) | 9,677 (16.4%) | -0.11 | 8,220 (15.1%) | 8,160 (15.0%) | 0.00 |
|---|---|---|---|---|---|---|
| Chronic liver disease | 4,934 (6.6%) | 4,700 (8.0%) | -0.05 | 4,057 (7.4%) | 4,087 (7.5%) | 0.00 |
| Asthma | 10,136 (13.6%) | 9,418 (16.0%) | -0.07 | 8,320 (15.2%) | 8,327 (15.3%) | 0.00 |
| Ischemic heart disease | 20,526 (27.5%) | 16,408 (27.9%) | -0.01 | 15,080 (27.6%) | 15,093 (27.7%) | 0.00 |
| Chronic obstructive pulmonary | | | | | | |
| disease | 16,838 (22.5%) | 14,000 (23.8%) | -0.03 | 12,732 (23.3%) | 12,806 (23.5%) | 0.00 |
| Malignancy | 18,107 (24.2%) | 15,987 (27.2%) | -0.07 | 14,290 (26.2%) | 14,308 (26.2%) | 0.00 |
| Drug or alcohol abuse or | | | | | | |
| dependence | 6,027 (8.1%) | 4,518 (7.7%) | 0.01 | 4,239 (7.8%) | 4,250 (7.8%) | 0.00 |
| Venous thromboembolism | 3,540 (4.7%) | 3,109 (5.3%) | -0.03 | 2,760 (5.1%) | 2,793 (5.1%) | 0.00 |

#### 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>7</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease.

#### 10. References

- 1. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 2. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **3.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* May 2012;21 Suppl 2:69-80.
- **4.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- 5. AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. Comp Effect Res 2013;3:11-20.
- **6.** Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- 7. Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.

| # | Implementation in routine care | |
|---|---|---|
| | | EXPOSURE vs. COMPARISON |
| | Methotrexate vs Hydroxychloroquine | INCLUCION CRITERIA |
| | No prior use of methotrexate or | INCLUSION CRITERIA Depending on the comparison group, we will require new-use (defined as no use anytime prior to index date) of |
| 1 | hydroxychloroquine | methotrexate and hydroxychloroquine |
| 2 | Sufficient enrollment | Medicare Part A, B, and D enrollment with no HMO coverage for 365 days prior to and on the cohort entry date |
| | | EXCLUSION CRITERIA |
| | Prior history of dementia | Measured any time prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| | | ICD9 diagnosis – 046.1x, 290.xx (excluding 290.8), 291.2, 292.82, 294.1x, 294.2x, 331.0-331.2, 331.7, 331.82, 331.83, 333.4, 780.93, 797 ICD10 diagnosis – F01.xx-F03.xx, G30.xx-G31.85, R41.xx |
| 1 | | NDC brand name – ""ARICEPT", "ARICEPT ODT", "EXELON", "NAMENDA", "NAMENDA XR", "NAMZARIC", "RAZADYNE", "RAZADYNE ER", or "REMINYL" |
| | | NDC generic name – "DONEPEZIL HCL", "GALANTAMINE HBR", "MEMANTINE HCL", "MEMANTINE HCL/DONEPEZIL HCL", "RIVASTIGMINE", or "RIVASTIGMINE TARTRATE" |
| | No prior history of rheumatoid arthritis | Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| 2 | | ICD9 diagnosis – 714.xx<br>ICD10 diagnosis – M05.xx, M06.xx, M08.xx, M12.xx |
| | Nursing home admission | Measured 365 days prior to drug initiation – |
| 3 | | MEDPAR - Short Stay/Long Stay/SNF Indicator Code – N = SNF Stay (Prvdr3 = 5, 6, U, W, Y, or Z) |
| | Prior history of DMARD use | Measured 365 days prior to drug initiation – |
| | | HCPCS procedure code – J0135, C9249, J0717, J0718, J1438, J1602, J1745, C9230, J0129, C9264, J3262, J1600, J9310 |
| 4 | | NDC brand name — "HUMIRA", "CIMZIA", "ENBREL", "SIMPONI", "SIMPONI ARIA", "REMICADE", "ORENCIA", "ACTEMRA", "XELJANZ", "RIDAURA", "AZASAN", "AZATHIOPRINE", "AZATHIOPRINE SODIUM", "IMURAN", "CYCLOSPORINE", "CYCLOSPORINE MODIFIED", "GENGRAF", "NEORAL" "RESTASIS", "SANDIMMUNE", "SANGCYA", "CYCLOPHOSPHAMIDE", "CYCLOPHOSPHAMIDE MONOHYDRATE", "CYTOXAN", "CYTOXAN LYOPHILIZED", "NEOSAR", "NEOSAR FOR INJECTION", "AUROLATE", "GOLD SODIUM THIOMALATE", "MYOCHRYSINE", "ARAVA", "LEFLUNOMIDE", "AZULFIDINE", "S.A.S500", "SULFA DYNE", "SULFASALAZINE", "SULFASALAZINE DR", "SULFAZINE EC", "KINERET", "RITUXAN" |
| | | NDC generic name — "ADALIMUMAB", "CERTOLIZUMAB PEGOL", "ETANERCEPT", "GOLIMUMAB", "INFLIXIMAB", "ABATACEPT", "ABATACEPT/MALTOSE", "TOCILIZUMAB", "TOFACITINIB CITRATE", "AURANOFIN", "AZATHIOPRINE", "AZATHIOPRINE SODIUM", "CYCLOSPORINE", "CYCLOSPORINE, MODIFIED", "CYCLOPHOSPHAMIDE", "GOLD SODIUM THIOMALATE", "LEFLUNOMIDE", "SULFASALAZINE", "ANAKINRA", "RITUXIMAB" |

| Covariate list | |
|---|---|
| | Potential confounders |
| Category | ICD-9 |
| | Age |
| | Gender |
| | Race |
| Demographics | Region |
| | Calendar year of index date |
| | Low income subsidy |
| | Diabetes |
| | Obesity |
| | Hypertension |
| | Coronary artery disease |
| Dementia risk factors | Depression |
| | Anxiety |
| | Bipolar disorder |
| | Schizophrenia |
| | Smoking |
| | Mammography |
| | Colonoscopy |
| | Fecal occult blood test |
| Lifestyle factors and markers for healthy behavior | Influenza vaccination |
| | Pneumococcal vaccination |
| | Herpes zoster vaccination |
| | BMD test |
| | Number of distinct generic agents |
| | Number of emergency room visits |
| | Number of outpatient visits |
| Haddan (Pratta and a | Number of hospitalizations |
| Healthcare utilization measures | Number of physician office visits |
| | Number of rheumatologist visits |
| | Number of CRP tests ordered |
| | Number of serum creatinine tests ordered |
| | Composite frailty score |
| | Osteoporosis |
| Frailty markers | Fractures |
| rancy markets | Falls |
| | Use of supplemental oxygen |
| | A combined comorbidity score |
| RA-specific como | orbidities |
| | Lithium |
| | Anti-epileptic mood stabilizers |
| | Anti-epileptics (other than mood stabilizers) |

| | Atypical antipsychotics |
|---|---|
| | Benzodiazepines |
| | SNRIs |
| | SSRIs |
| | TCAs |
| | Typical antipsychotics |
| | Anticoagulants |
| Comedications | Antiplatelet agents |
| | Angiotensin II receptor blockers |
| | Angiotensin converting enzyme inhibitors |
| | Beta blockers |
| | Calcium channel blockers |
| | Diuretics |
| | Nitrates |
| | Lipid lowering drugs |
| | Non-insulin diabetes medications |
| | Insulin |
| | Antidepressants |
| | инисрессовно |
| | Number of biologic DMARDs |
| | Number of nonbiologic DMARDs |
| | Use of other nonbiologic DMARDs |
| | Methotrexate |
| | Hydroxychloroguine |
| | Leflunomide |
| | Sulfasalazine |
| Nonbiologics | Anakinra |
| | Auranofin |
| | Azathioprine |
| | Cyclosporine |
| | Cyclosphosphamide |
| | Gold sodium thiomalate |
| | NSAID/COXIB |
| | Opioids |
| | Glucocorticoids |
| | Atrial fibrillation |
| | Coronary artery disease |
| | Heart failure |
| | Stroke or TIA |
| | Peripheral vascular disease |
| | Hypertension |
| | Diabetes |
| | Hyperlipidemia |
| Com orbid conditions | |
| Com orbid conditions | Hyperlipidemia Renal dysfunction Chronic liver disease |
| Com orbid conditions | Renal dysfunction |

# Appendix A

| COPD |
|-------------------------------------|
| Malignancy |
| Drug or alcohol abuse or dependence |
| VTE |

## Appendix A Demographics

| Calendar year of index date |
|-----------------------------|
| Year |
| 2007 |
| 2008 |
| 2009 |
| 2010 |
| 2011 |
| 2012 |
| 2013 |
| 2014 |
| 2015 |
| 2016 |
| 2017 |

#### Low income subsidy

https://www.cms.gov/Medicare/Eligibility-and-

 $\underline{\textbf{Enrollment/LowIncSubMedicarePresCov/Downloads/StateLISGuidance021009.pd}}$ 

£

#### Diabetes


Obesity


### Prescriptions

Orlistat
Sibutramine
Phentermine
Benzphetamine
Phendimetrazine
Diethylpropion

Hypertension

| Hypertension | | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
| I10 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| I10 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| I10 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| I160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| l161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| I169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| I110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| I110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart |
| I110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, malignant, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | kidney disease stage I through stage IV, or unspecified |
| | | disease | |
| I120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| l129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and with chronic kidney disease stage V |
| | | stage renal disease | or end stage renal disease |

| I1310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
|---|---|---|---|
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end | heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| 1150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| l151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| l152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| 1158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| 1159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

Coronary artery disease


| equent ST elevation (STEMI) myocardial infarction of | Acute myocardial infarction of inferolateral wall, initial |
|---|---|
| or wall | episode of care |
| evation (STEMI) myocardial infarction involving other ary artery of inferior wall | Acute myocardial infarction of inferolateral wall, subsequent episode of care |
| evation (STEMI) myocardial infarction involving right | Acute myocardial infarction of inferoposterior wall, episode of care unspecified |
| evation (STEMI) myocardial infarction involving right | Acute myocardial infarction of inferoposterior wall, initial episode of care |
| equent ST elevation (STEMI) myocardial infarction of | Acute myocardial infarction of inferoposterior wall, initial |
| or wall<br>evation (STEMI) myocardial infarction involving right | episode of care Acute myocardial infarction of inferoposterior wall, |
| ary artery evation (STEMI) myocardial infarction involving other | subsequent episode of care Acute myocardial infarction of other inferior wall, episode of |
| evation (STEMI) myocardial infarction involving other | care unspecified<br>Acute myocardial infarction of other inferior wall, initial |
| ary artery of inferior wall equent ST elevation (STEMI) myocardial infarction of | episode of care Acute myocardial infarction of other inferior wall, initial |
| or wall evation (STEMI) myocardial infarction involving other | episode of care Acute myocardial infarction of other inferior wall, |
| ary artery of inferior wall | subsequent episode of care |
| evation (STEMI) myocardial infarction involving other | Acute myocardial infarction of other lateral wall, episode of care unspecified |
| evation (STEMI) myocardial infarction involving other | Acute myocardial infarction of other lateral wall, initial episode of care |
| equent ST elevation (STEMI) myocardial infarction of | Acute myocardial infarction of other lateral wall, initial episode of care |
| evation (STEMI) myocardial infarction involving other | Acute myocardial infarction of other lateral wall, |
| evation (STEMI) myocardial infarction involving other | subsequent episode of care True posterior wall infarction, episode of care unspecified |
| evation (STEMI) myocardial infarction involving other | True posterior wall infarction, initial episode of care |
| equent ST elevation (STEMI) myocardial infarction of | True posterior wall infarction, initial episode of care |
| evation (STEMI) myocardial infarction involving other | True posterior wall infarction, subsequent episode of care |
| T elevation (NSTEMI) myocardial infarction | Subendocardial infarction, episode of care unspecified |
| | Subendocardial infarction, initial episode of care |
| | Subendocardial infarction, initial episode of care |
| | Subendocardial infarction, subsequent episode of care |
| evation (STEMI) myocardial infarction involving other | Acute myocardial infarction of other specified sites, episode of care unspecified |
| evation (STEMI) myocardial infarction involving left | Acute myocardial infarction of other specified sites, initial episode of care |
| evation (STEMI) myocardial infarction involving other | Acute myocardial infarction of other specified sites, initial episode of care |
| equent ST elevation (STEMI) myocardial infarction of | Acute myocardial infarction of other specified sites, initial |
| evation (STEMI) myocardial infarction involving other | episode of care Acute myocardial infarction of other specified sites, |
| evation (STEMI) myocardial infarction of unspecified | subsequent episode of care Acute myocardial infarction of unspecified site, episode of |
| evation (STEMI) myocardial infarction of unspecified | care unspecified Acute myocardial infarction of unspecified site, initial |
| equent ST elevation (STEMI) myocardial infarction of | episode of care Acute myocardial infarction of unspecified site, initial |
| ecified site<br>evation (STEMI) myocardial infarction of unspecified | episode of care Acute myocardial infarction of unspecified site, subsequent |
| -Design 10 | episode of care |
| | LongDeslCD9 |
| osclerotic heart disease of native coronary artery out angina pectoris | Coronary atherosclerosis of unspecified type of vessel, native or graft |
| | evation (STEMI) myocardial infarction involving other ary artery of inferior wall evation (STEMI) myocardial infarction involving right ary artery evation (STEMI) myocardial infarction involving right ary artery quent ST elevation (STEMI) myocardial infarction involving right ary artery quent ST elevation (STEMI) myocardial infarction involving right ary artery evation (STEMI) myocardial infarction involving other ary artery of inferior wall evation (STEMI) myocardial infarction involving other ary artery of inferior wall evation (STEMI) myocardial infarction involving other ary artery of inferior wall evation (STEMI) myocardial infarction involving other ary artery of inferior wall evation (STEMI) myocardial infarction involving other ary artery of inferior wall evation (STEMI) myocardial infarction involving other evation (STEMI) myocardial infarction of unspecified evation (STEMI) myocardial infarction of unspecified evation (STEMI) myocardial infarction of unspecified evation (STEMI) myocardial infarction of unspecified evation (STEMI) myocardial infarction of unspecified evation (STEMI) myocardial infarcti |


Depression


#### Anxiety


#### Bipolar disorder


# Appendix A Dementia risk factors


#### Schizophrenia


#### Smoking


CPT codes

99406

99407

G0436

G0437

G9016

S9453

S4995

G9276

G9458

1034F

4001F

4004F

OR dispensing of: At least one nicotine or varenicline prescription

#### Mammography


Colonoscopy


**CPT**45378
45379

50

Appendix A Lifestyle factors and markers for healthy behavior

| 45380 |
|-------|
| 45381 |
| 45382 |
| 45383 |
| 45384 |
| 45385 |
| 45386 |
| 45387 |
| 45388 |
| 45389 |
| 45390 |
| 45391 |
| 45392 |
| HCPCS |
| G0105 |
| G0121 |

### Fecal occult blood test


### Influenza vaccination


#### Pneumococcal vaccination


Appendix A Lifestyle factors and markers for healthy behavior

| 90670 |
|-------|
| 90732 |

### Herpes zoster vaccination

| • |
|-------|
| CPT |
| 90376 |
| 90750 |

#### BMD test

| CPT |
|-------|
| 76070 |
| 76075 |
| 76076 |
| 76977 |
| 77080 |
| 77085 |

#### Healthcare utilization measures

#### Number of generic medications

NDC generic drug name has any value

If multiple events on a single day, the value is measured as combined values.

#### Number of ED visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99281 | 99282 | 99283 | 99284 | 99285 | 99288 |

#### Number of outpatient visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99450 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99455 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99456 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99499 |
| 99213 | 99271 | 99357 | 99391 | 99402 | |

#### Number of hospitalizations

The occurrence of MEDPAR with the following attributes:

Inpatient admission type code exists

The occurrence of carrier claims with the following attributes:

20 = Non swing bed SNF claim

30 = Swing bed SNF claim

50 = Hospice claim

60 = Inpatient claim

61 = Inpatient 'full-encounter' claim

#### Number of PCP visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

01 = General practice

08 = Family practice

11 = Internal medicine

84 = Preventive medicine (eff 5/92)

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99429 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99450 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99455 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99456 |
| 99213 | 99271 | 99357 | 99391 | 99402 | 99499 |

#### Number of rheumatologist visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

66 = Rheumatology (eff 5/92) Note: during 93/94 DMERC also used this to mean medical supply company with respiratory therapist

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99000 | 99141 | 99249 | 99347 | 99450 | 99603 |
| 99001 | 99142 | 99250 | 99348 | 99454 | 99604 |
| 99002 | 99143 | 99251 | 99349 | 99455 | 99605 |
| 99003 | 99144 | 99252 | 9934S | 99456 | 99606 |
| 99004 | 99145 | 99253 | 99350 | 99460 | 99607 |
| 99005 | 99148 | 99254 | 99351 | 99461 | 99615 |
| 99006 | 99149 | 99255 | 99352 | 99462 | 99649 |
| 99010 | 09915 | 99256 | 99353 | 99463 | 99675 |
| 99011 | 99150 | 9925S | 99354 | 99464 | 99684 |
| 99012 | 99160 | 99261 | 99355 | 99465 | 99700 |
| 99014 | 99163 | 99262 | 99356 | 99466 | 99703 |
| 99015 | 99166 | 99263 | 99357 | 99467 | 99707 |
| 99020 | 99170 | 99270 | 99358 | 99468 | 99713 |
| 99023 | 99171 | 99271 | 99359 | 99469 | 99714 |

| 99024 | 00172 | 00272 | 00350 | 00470 | 00717 |
|-------|-------|-------|-------|-------|-------|
| | 99172 | 99272 | 9935D | 99470 | 99717 |
| 99025 | 99173 | 99273 | 99360 | 99471 | 99732 |
| 99026 | 99174 | 99274 | 99361 | 99472 | 99736 |
| 99027 | 99175 | 99275 | 99362 | 99475 | 99762 |
| 99028 | 99178 | 99280 | 99363 | 99476 | 99770 |
| 99032 | 99183 | 99281 | 99364 | 99477 | 99772 |
| 99035 | 99184 | 99282 | 99365 | 99478 | 99776 |
| 99038 | 99185 | 99283 | 99366 | 99479 | 99780 |
| 99039 | 99186 | 99284 | 99367 | 99480 | 99799 |
| 99040 | 99188 | 99285 | 99368 | 99481 | 9979A |
| 99041 | 99190 | 99286 | 99371 | 99482 | 99801 |
| 99042 | 99191 | 99287 | 99372 | 99485 | 99802 |
| 99045 | 99192 | 99288 | 99373 | 99486 | 99803 |
| 99047 | 99195 | 99289 | 99374 | 99487 | 99806 |
| 99048 | 99199 | 99290 | 99375 | 99488 | 99810 |
| 99049 | 99200 | 99291 | 99376 | 99489 | 99811 |
| 99050 | 99201 | 99292 | 99377 | 99490 | 99814 |
| 99051 | 99202 | 99293 | 99378 | 99495 | 99821 |
| 99052 | 99203 | 99294 | 99379 | 99496 | 99833 |
| 99053 | 99204 | 99295 | 99380 | 99497 | 99840 |
| 99054 | 99205 | 99296 | 99381 | 99498 | 99841 |
| 99056 | 99206 | 99297 | 99382 | 99499 | 99881 |
| 99058 | 99207 | 99298 | 99383 | 99500 | 99894 |
| 99060 | 99208 | 99299 | 99384 | 99501 | 99897 |
| 99063 | 99209 | 9930 | 99385 | 99502 | 99899 |
| 99065 | 9920A | 99300 | 99386 | 99503 | 99901 |
| 99070 | 9920X | 99301 | 99387 | 99504 | 99902 |
| 99071 | 09921 | 99302 | 99391 | 99505 | 99907 |
| 99072 | 99210 | 99303 | 99392 | 99506 | 99910 |
| 99074 | 99211 | 99304 | 99393 | 99507 | 99912 |
| 99075 | 99212 | 99305 | 99394 | 99508 | 99913 |
| 99076 | | | | | |
| | 99213 | 99306 | 99395 | 99509 | 99914 |
| 99078 | 99214 | 99307 | 99396 | 99510 | 99919 |
| 99079 | 99215 | 99308 | 99397 | 99511 | 99920 |
| 9907B | 99216 | 99309 | 99399 | 99512 | 99921 |
| 9907E | 99217 | 99310 | 99400 | 99513 | 99925 |
| 99080 | 99218 | 99311 | 99401 | 99514 | 99931 |
| 99081 | 99219 | 99312 | 99402 | 99523 | 99940 |
| 99082 | 9921F | 99313 | 99403 | 99530 | 99941 |
| 99089 | 9921G | 99315 | 99404 | 99539 | 99942 |
| 99090 | 9921S | 99316 | 99406 | 99551 | 99943 |
| 99091 | 99220 | 99317 | 99407 | 99552 | 99949 |
| 99097 | 99221 | 99318 | 99408 | 99553 | 99959 |
| 99099 | 99222 | 99321 | 99409 | 99554 | 99960 |
| 990ST | 99223 | 99322 | 9940A | 99555 | 99961 |
| 99100 | 99224 | 99323 | 99411 | 99556 | 99968 |
| 99101 | 99225 | 99324 | 99412 | 99557 | 99970 |
| 99102 | 99226 | 99325 | 99420 | 99558 | 99989 |
| 99102 | 99227 | 99326 | 99429 | 99559 | 09999 |
| 99110 | 99230 | 99327 | 9942G | 99560 | 99990 |
| 99111 | 99231 | 99328 | 99431 | 99561 | 99991 |
| 99112 | 99232 | 99331 | 99432 | 99562 | 99992 |
| 99113 | 99233 | 99332 | 99433 | 99563 | 99993 |
| 99115 | 99234 | 99333 | 99435 | 99564 | 99994 |
| 99116 | 99235 | 99334 | 99436 | 99565 | 99995 |
| 99119 | 99236 | 99335 | 99438 | 99566 | 99996 |
| 99120 | 99238 | 99336 | 99440 | 99567 | 99997 |
| 99121 | 99239 | 99337 | 99441 | 99568 | 99998 |
| 99123 | 99241 | 99339 | 99442 | 99569 | 99999 |
| 99124 | 99242 | 99340 | 99443 | 99580 | 9999G |
| 99125 | 99243 | 99341 | 99444 | 99588 | 9999V |
| 09913 | 99244 | 99342 | 99446 | 99593 | 99Z14 |
| 99135 | 99245 | 99343 | 99447 | 99600 | |
| 09914 | 99246 | 99344 | 99448 | 99601 | |
| | l | | | | |
| 99140 | 99248 | 99345 | 99449 | 99602 | |



## Appendix A Healthcare utilization measures

| 86140 | 86141 |
|-------|-------|

#### Number of serum creatinine tests

| CPT | |
|-------|-------|
| 80048 | 80054 |
| 80049 | 80069 |
| 80053 | 82565 |

#### Frailty Score for Claims Data

Kim DH. Schneeweiss S. Glynn RJ. Lipsitz LA. Rockwood K. Avorn J. Measuring frailty in Medicare data: Development and validation of a claims-based frailty index. Journals of Gerontology: Medical Sciences 2018;73(7):980-87.

Codes used for each component of the frailty score

| Codes used for each component of the fra<br>Condition | ICD9 Dx | ICD10 Dx | Coefficient |
|---|---|---|---|
| Intercept | | | 0.10288 |
| Intestinal infectious diseases | 001-009 | A00-A09 (exclude A02.1) | 0.00582 |
| Other and unspecified effects of external causes | 990-995 | A02.1, A22.7, A26.7, A32.7, A40, A41, A42.7, A45.8, B37.7, R65, T33, T34, T36-T50, T66-T78, T88 | 0.0085 |
| Other bacterial diseases | 030-041 | A30-A39; A42-A49 (exclude A32.7,A42.7,A45) | 0.01188 |
| Mycoses | 110-118 | B35-B49 (exclude B37.7) | 0.00831 |
| Malignant neoplasm of other and unspecified sites | 190-199 | C69-C80 | 0.00797 |
| Organic psychotic conditions | 290-294 | D01, D03, F02, F04, F05, F06, F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.122, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.982, F19.999, F19.94, F19.950, F19.951, F19.96, F19.97, F19.99 | 0.04745 |
| Benign neoplasms | 210-229 | D10-D36 | -0.00513 |
| Neoplasms of uncertain behavior | 235-238 | D37-D48 | -0.00061 |
| Other and unspecified anemias | 285 | D62, D64 | 0.0085 |
| Purpura and other hemorrhagic conditions | 287 | D69 | -0.00804 |
| Diseases of white blood cells | 288 | D70, D71, D72, D76 | -0.0068 |
| Other metabolic and immunity disorders | 270-279 | D80-D84, D89, E65-E68, E70-E88, M10 (exclude E75.02, E75.19, E75.23, E75.25, E75.29, E75.4) | -0.00564 |
| Disorders of thyroid gland | 240-246 | E00-E07 | 0.00439 |
| Diseases of other endocrine glands | 250-259 | E08-E16,E20-E35 | 0.01078 |
| Hereditary and degenerative diseases of the central nervous system | 330-337 | E75.02, E75.19, E75.23, E75.25, E75.29, E75.4, F84.2, G10, G11, G12, G20, G21.0, G23, G24, G25, G30.9, G31, G80.3, G90, G91, G93.7, G93.89, G93.9, G94, G95, G99.2 | 0.01078 |

| Neurotic Disorders, Personality<br>Disorders, And Other Nonpsychotic<br>Mental Disorders | 300-316 | F07, F09, F32.9, F40-F44, F48, F54, F60, F64-F66, F68, F10-F19, F45.8, F45.9, F50, F51, F63.3, F80-F82, F88-F91, F93-F95, F98, R45.1, R48.0 (exclude F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F14.982, F14.988, F15.122, F15.159, F15.180, F15.181, F15.182, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.921, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, | 0.01353 |
|---|---|---|---|
| Other psychoses | 295-299 | F20, F22-F25, F28-F34, F39, F44.89, F84 (exclude F84.2, F32.9) | 0.02112 |
| Other disorders of the central nervous system | 340-349 | G35, G37, G40, G43, G47.4, G80-G83, G92, G93.0-G93.2, G93.4-G93.6, G96-G97, G98.8 (exclusion G80.3 ) | 0.04031 |
| Disorders of the peripheral nervous system | 350-359 | G60-G65 | 0.00338 |
| Disorders of the eye and adnexa | 360-379 | H00-H59 (exclude H54.7) | -0.00061 |
| Hypertensive disease | 401-405 | 110-116 | 0.0174 |
| Ischemic heart disease | 410-414 | 120-125 | 0.0192 |
| Other forms of heart disease | 420-429 | 130-152 | 0.01989 |
| Cerebrovascular disease | 430-438 | 160-169 | -0.00046 |
| Diseases of arteries, arterioles, and capillaries | 440-448 | 170-179 | 0.00106 |
| Diseases of veins and lymphatics, and other diseases of circulatory system | 451-459 | 180-189;195-199 | 0.01234 |
| Pneumonia and influenza | 480-487 | J09-J18 | 0.01185 |
| Other diseases of the upper respiratory tract | 470-478 | 130-139 | -0.0052 |
| Chronic obstructive pulmonary disease and allied conditions | 490-496 | J40-J45,J47,J67 | 0.01295 |
| Diseases of oral cavity, salivary glands, and jaws | 520-529 | K00-K14 | 0.00261 |
| Diseases of esophagus, stomach, and duodenum | 530-537 | K20-K31 | 0.0005 |
| Hernia of abdominal cavity | 550-553 | K40-K46 | 0.00388 |
| Infections of skin and subcutaneous tissue | 680-686 | L00-L08 | 0.00561 |
| Other inflammatory conditions | 690-698 | L10-L49, L51-L59 | -0.00053 |
| Arthropathies and related disorders | 710-719 | M00-M02, M04, M05-M09 M11-M14, M15-M19, M20-M25, M30-M36 (excluded M35.3) | 0.01408 |
| Rheumatism, excluding the back | 725-729 | M35.3, M60-M79,R25.2,R29.8x | 0.00021 |
| Dorsopathies | 720-724 | M40-M54 | 0.00984 |

| Osteopathies, chondropathies, and acquired musculoskeletal deformities | 730-739 | M80-M85, M86-M90, M91-M95, M99 | 0.00389 |
|---|---|---|---|
| Nephritis, nephrotic syndrome, and nephrosis | 580-589 | N00-N05, N08,N17,N18, N25, N26,N27 | 0.01047 |
| Other diseases of urinary system | 590-599 | N30-N39 | 0.01062 |
| Diseases of male genital organs | 600-608 | N40-N53 | -0.02131 |
| Congenital anomalies in urinary system | 753 | Q60-Q64 | -0.00836 |
| Congenital anomalies in musculoskeletal system | 754-756 | Q65-Q79 | 0.00073 |
| Symptoms | 780-789 | R00-R39, R50-R63 (exclude R09.1, R09.2,R13,R25.2,R29.8,R51, R52) | 0.00593 |
| III-defined and unknown causes of morbidity and mortality | 797-799 | R09.1, R09.2,R41.8x,R68.13,R68.82, R64,R69,R99 | 0.01119 |
| Nonspecific abnormal findings | 790-796 | R70-R97 | -0.00231 |
| Contusion with intact skin surface | 920-924 | \$00.93, \$10.93, \$00.10-\$00.12, \$05.10-\$05.12, \$05.90-\$05.92, \$20.00-\$20.02, \$20.20-\$20.22, \$30.0-\$30.3, T14.8-T14.9, \$40.01-\$40.02, \$50.0-\$50.1, \$60.0-\$60.2, \$70.0-\$70.1, \$80.0-\$80.1, \$90.0-\$90.3 | 0.01074 |
| Open wound of lower limb | 890-897 | S81 | 0.02042 |
| Persons with a condition influencing their health status | V40-V49 | F48.9, F52.9, F69, F81.9, H54.7, H93.9x, J95.850, M96.0, R13.10, R43.9, R46.8x, R47.89, R68.89, Z48.22-Z48.298, Z66, Z73.82, Z74.0x, Z76.82, Z78.x, Z86.59, Z87.898, Z89.0x (excluding 789.52x), 790.x (excluding (Z90.41x. Z90.71x), 791.15, 791.83, 792.82, 793.x-795.x, 796.3x-Z96.9, 797.x-799.x (excluding 798.5x, 795.87x) | 0.00191 |
| Persons without reported diagnosis encountered during examination and investigation of individuals and populations | V70-V82 | Z00-Z13 | -0.01208 |
| Persons with potential health hazards related to communicable diseases | V01-V09 | Z20-Z29 | -0.00189 |
| Persons encountering health services for specific procedures and aftercare | V50-V59 | Z40-Z53, Z79 (exclude Z48.280, Z48.23, Z48.24, Z48.288, Z48.298 , Z48.22, Z48.290) | 0.00118 |

| Condition | CPT Code | Coefficient |
|---|---|---|
| Office/other outpatient visit – established patient | 99214 | 0.00149 |
| Hospital care – initial | 99222 | 0.0017 |
| Office consultation | 99242 | -0.00094 |
| Office consultation | 99245 | 0.00169 |
| Nursing facility care – subsequent | 99308 | 0.01389 |
| Preventive medicine services | 99381-99429 | -0.00712 |
| Anesthesia – head | 00100-00222 | -0.00049 |
| Anesthesia – neck | 00300-00352 | 0.00614 |
| Anesthesia – intrathoracic | 00500-00580 | -0.01568 |
| Anesthesia – lower abdomen | 00800-00882 | -0.01053 |
| Anesthesia – knee and popliteal area | 01320-01444 | -0.01215 |
| Surgery – respiratory system | 30000-32999 | -0.00129 |
| Surgery – female genital system | 56405-58999 | 0.00327 |
| Surgery – nervous system | 61000-64999 | 0.00843 |
| Radiology – nuclear medicine | 78000-79999 | -0.00301 |
| Therapeutic drug assays | 80150-80299 | 0.00789 |
| Cytopathology | 88104-88199 | -0.01082 |
| Surgical pathology | 88300-88399 | -0.00427 |

| Medicine – Ophthalmology | 92002-92499 | -0.00295 |
|----------------------------------------------------|-------------|----------|
| Medicine – Cardiovascular | 92950-93799 | -0.00046 |
| Medicine – Noninvasive vascular diagnostic studies | 93875-93990 | -0.00828 |
| Allergy and clinical immunology | 95004-95199 | -0.0084 |
| Physical medicine and rehabilitation | 97001-97799 | -0.00012 |
| Chiropractic manipulative treatment | 98940-98943 | -0.01426 |
| Special services, procedures and reports | 99000-99091 | 0.00127 |

| Condition | HCPCS Code | Coefficient |
|---|---|---|
| Transportation services including ambulance | A0021-A0999 | 0.01022 |
| Other supplies including diabetes supplies and contraceptives | A4244-A4290 | 0.0236 |
| Diabetic footwear | A5500-A5513 | 0.02375 |
| Breathing aids | A7000-A7046 | 0.00947 |
| Administrative, miscellaneous and experimental | A9150-A9999 | -0.00167 |
| Walking aids and attachments | E0100-E0159 | 0.02821 |
| Hospital beds and associated supplies | E0250-E0373 | 0.08649 |
| Oxygen delivery systems and related supplies | E0424-E0486 | 0.00665 |
| Humidifiers and nebulizers with related equipment | E0550-E0601 | 0.00385 |
| Wheelchair or transport chair and related accessories | E0950-E1298,<br>E2201-E2294,<br>E2300-E2399,<br>E2601-E2621 | 0.00805 |
| Accessories for oxygen delivery devices | E1353-E1406 | 0.02702 |
| Vaccine administration | G0008-G0010 | -0.00158 |
| Screening examinations and disease management training | G0101-G0124 | -0.01136 |
| Drugs, administered by injection | J0120-J7130 | 0.00664 |
| Inhalation solutions | J7608-J7684 | 0.00412 |
| Wheelchairs, components, and accessories | K0001-K0462,<br>K0669 | 0.07802 |

Osteoporosis

| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDesICD9 |
|---|---|---|---|
| M810 | 73300 | Age-related osteoporosis without current pathological | Osteoporosis, unspecified |
| | | fracture | |
| M810 | 73301 | Age-related osteoporosis without current pathological | Senile osteoporosis |
| | | fracture | |
| M818 | 73302 | Other osteoporosis without current pathological fracture | Idiopathic osteoporosis |
| M818 | 73303 | Other osteoporosis without current pathological fracture | Disuse osteoporosis |
| M816 | 73309 | Localized osteoporosis [Lequesne] | Other osteoporosis |
| M818 | 73309 | Other osteoporosis without current pathological fracture | Other osteoporosis |


| encounter and extradural hemorrh consciousness S065X0A 80120 Traumatic subdural hemorrhage without loss of consciousness, initial encounter and extradural hemorrh | of skull with subarachnoid, subdural, |
|---|---|
| S065X0A 80120 Traumatic subdural hemorrhage without loss of consciousness, initial encounter and extradural hemorrh | nage unenecified state of |
| S065X0A 80120 Traumatic subdural hemorrhage without loss of consciousness, initial encounter and extradural hemorrh | lage, unspecified state of |
| consciousness, initial encounter and extradural hemorrh | af alvelles ithe authorization and authorization |
| | · |
| | nage, unspecified state of |
| consciousness | |
| S066X0A 80120 Traumatic subarachnoid hemorrhage without loss of Closed fracture of base | of skull with subarachnoid, subdural, |
| consciousness, initial encounter and extradural hemorrh | nage, unspecified state of |
| consciousness | |
| S02109A 80121 Fracture of base of skull, unspecified side, initial encounter Closed fracture of base | of skull with subarachnoid, subdural, |
| | nage, with no loss of consciousness |
| | iage, men no ross er consciousness |
| S064X0A 80121 Epidural hemorrhage without loss of consciousness, initial Closed fracture of base | of skull with subarachnoid, subdural, |
| | nage, with no loss of consciousness |
| and extradular nemorn | lage, with no loss of consciousness |
| COCCYOA 20121 Traumatic subdural homographore without loss of Closed fracture of hose | of clault with cubora shootd cubdural |
| | of skull with subarachnoid, subdural, |
| consciousness, initial encounter and extradural hemorrh | nage, with no loss of consciousness |
| | of skull with subarachnoid, subdural, |
| consciousness, initial encounter and extradural hemorrh | nage, with no loss of consciousness |
| | of skull with subarachnoid, subdural, |
| for closed fracture and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| S064X1A 80122 Epidural hemorrhage with loss of consciousness of 30 minutes Closed fracture of base | of skull with subarachnoid, subdural, |
| or less, initial encounter and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| | of skull with subarachnoid, subdural, |
| | nage, with brief [less than one hour] |
| loss of consciousness | lage, with bire fless than one floar |
| | af alvelles ith as because the side as the decide |
| | of skull with subarachnoid, subdural, |
| | nage, with brief [less than one hour] |
| loss of consciousness | |
| S065X2A 80122 Traumatic subdural hemorrhage with loss of consciousness of Closed fracture of base | of skull with subarachnoid, subdural, |
| 31 minutes to 59 minutes, initial encounter and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| S066X1A 80122 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base | of skull with subarachnoid, subdural, |
| consciousness of 30 minutes or less, initial encounter and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| S066X2A 80122 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base | of skull with subarachnoid, subdural, |
| <u> </u> | nage, with brief [less than one hour] |
| | lage, with bire fless than one hoar] |
| loss of consciousness S03100A 90133 Eracture of base of skull unspecified side initial ensembles. Closed fracture of base | of ckull with subarasbasid subdivis |
| | of skull with subarachnoid, subdural, |
| | nage, with moderate [1-24 hours] los |
| of consciousness | |
| | of skull with subarachnoid, subdural, |
| hours 59 minutes, initial encounter and extradural hemorrh | nage, with moderate [1-24 hours] los |
| of consciousness | |
| S064X4A 80123 Epidural hemorrhage with loss of consciousness of 6 hours to Closed fracture of base | of skull with subarachnoid, subdural, |
| 24 hours, initial encounter and extradural hemorrh | nage, with moderate [1-24 hours] los |
| of consciousness | |
| | of skull with subarachnoid, subdural, |
| - 2002/201 - COTES - FILAMINATIC SAPARIAL HOLLIGIEE WITH 1033 OF COLISCIONSTICAS OF ICHOSEN HACELIE OF DATE | nage, with moderate [1-24 hours] loss |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh | |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness | of clault with cubarachasid subdiving |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of Closed fracture of base of the consciousness of Closed fracture of the consciousness of Closed fracture of Closed fracture of Closed fracture of Closed fra | |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh | · |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh of consciousness | nage, with moderate [1-24 hours] los |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh of consciousness S066X3A 80123 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base of consciousness | nage, with moderate [1-24 hours] lost |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh of consciousness S066X3A 80123 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base of consciousness | of skull with subarachnoid, subdural, nage, with moderate [1-24 hours] loss of skull with subarachnoid, subdural, nage, with moderate [1-24 hours] loss |


# Appendix A Frailty markers


## Falls


## Appendix A Frailty markers

#### Combined Comorbidity Score for Claims Data

Gagne II, Glynn RI, Avorn I, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of Clinical Epidemiology 2011:64(7):749-59.

Sun JW. Rogers JR. Her Q. Welch EC. Panozzo CA. Toh S. Gagne JJ. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. Medical Care. 2017 Dec 1:55(12):1046-51.

Codes used for each ICD-10-CM and ICD-9-CM version of the combined comorbidity score


# Appendix A Frailty markers


BM, backward mapping; GEMs, General Equivalence Mappings; FBM, forward-backward mapping; ICD-9-CM, International Classification of Diseases, 9<sup>th</sup> Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification

#### Lithium

| NDC Generic Name | |
|-------------------|------------------------------|
| LITHIUM ASPARTATE | LITHIUM CITRATE |
| LITHIUM CARBONATE | LITHIUM CITRATE TETRAHYDRATE |

#### Anti-epileptic mood stabilizers

| NDC Generic Name | |
|-------------------|---------------------------------------------------|
| CARBAMAZEPINE | OXCARBAZEPINE |
| DIVALPROEX SODIUM | VALPROIC ACID |
| LAMOTRIGINE | VALPROIC ACID (AS SODIUM SALT) (VALPROATE SODIUM) |

#### Anti-epileptic non-mood stabilizers

| Anti epitepite non mood stabilizers | |
|-------------------------------------|---------------|
| NDC Generic Name | |
| RUFINAMIDE | LACOSAMIDE |
| VIGABATRIN | ETHOSUXIMIDE |
| EZOGABINE | FELBAMATE |
| TIAGABINE HCL | LEVETIRACETAM |
| PHENYTOIN | TOPIRAMATE |
| ZONISAMIDE | PHENOBARBITAL |
| PRIMIDONE | GABAPENTIN |
| PREGABALIN | |

#### Atypical antipsychotics

| NDC Generic Name | |
|----------------------|---------------------|
| ZIPRASIDONE MESYLATE | ARIPIPRAZOLE |
| PALIPERIDONE | OLANZAPINE |
| ZIPRASIDONE HCL | RISPERIDONE |
| CLOZAPINE | QUETIAPINE FUMARATE |

#### Benzodiazepines

| 201120414120 | |
|-------------------------|----------------|
| NDC Generic Name | |
| ALPRAZOLAM | FLURAZEPAM HCL |
| CHLORDIAZEPOXIDE | LORAZEPAM |
| CLOBAZAM | MIDAZOLAM |
| CLONAZEPAM | OXAZEPAM |
| CLORAZEPATE DIPOTASSIUM | QUAZEPAM |
| DIAZEPAM | TEMAZEPAM |
| ESTAZOLAM | TRIAZOLAM |

#### Serotonin-norepinephrine reuptake inhibitor

| NDC Generic Name | |
|--------------------------|---------------------|
| DESVENLAFAXINE | DULOXETINE HCL |
| DESVENLAFAXINE FUMARATE | VENLAFAXINE HCL |
| DESVENLAFAXINE SUCCINATE | LEVOMILNACIPRAN HCL |

#### Selective serotonin reuptake inhibitor

| NDC Generic Name | |
|---------------------------|-----------------------------------------|
| PAROXETINE MESYLATE | CITALOPRAM HYDROBROMIDE |
| FLUOXETINE | FLUOXETINE HCL |
| OLANZAPINE/FLUOXETINE HCL | SERTRALINE HCL |
| FLUVOXAMINE MALEATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.17 |
| ESCITALOPRAM OXALATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.8 |
| PAROXETINE HCL | VILAZODONE HCL |

#### Tricyclic antidepressants

| NDC Generic Name | |
|------------------------------------|--------------------------------|
| PROTRIPTYLINE HCL | DESIPRAMINE HCL |
| IMIPRAMINE PAMOATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| TRIMIPRAMINE MALEATE | NORTRIPTYLINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE HCL |
| AMOXAPINE | DOXEPIN HCL |
| CLOMIPRAMINE HCL | AMITRIPTYLINE HCL |

#### Typical antipsychotics

| NDC Generic Name | |
|------------------------|--------------------------------|
| FLUPHENAZINE ENANTHATE | THIOTHIXENE |
| LOXAPINE | FLUPHENAZINE HCL |
| PIMOZIDE | PERPHENAZINE/AMITRIPTYLINE HCL |

| MESORIDAZINE BESYLATE | TRIFLUOPERAZINE HCL |
|------------------------|---------------------|
| MOLINDONE HCL | CHLORPROMAZINE HCL |
| THIOTHIXENE HCL | HALOPERIDOL |
| FLUPHENAZINE DECANOATE | THIORIDAZINE HCL |
| PERPHENAZINE | |

#### Anticoagulants

| NDC Generic Name | |
|---|---|
| APIXABAN | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE |
| DABIGATRAN ETEXILATE MESYLATE | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE/PF |
| DALTEPARIN SODIUM, PORCINE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER |
| EDOXABAN TOSYLATE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER/PF |
| ENOXAPARIN SODIUM | HEPARIN SODIUM, PORCINE/PF |
| FONDAPARINUX SODIUM | RIVAROXABAN |
| HEPARIN SODIUM,BEEF | TINZAPARIN SODIUM, PORCINE |
| HEPARIN SODIUM, PORCINE | WARFARIN SODIUM |
| HEPARIN SODIUM, PORCINE IN 0.45 % SODIUM CHLORIDE | |

#### Antiplatelet agents

| Antiplatelet agents | |
|---|---|
| NDC Generic Name | |
| ABCIXIMAB | CILOSTAZOL |
| ASPIRIN | CINNAMEDRINE HCL/ASPIRIN/CAFFEINE |
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN | CLOPIDOGREL BISULFATE |
| ASPIRIN/ACETAMINOPHEN | CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE | CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM | CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM | DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE | DIHYDROCODEINE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN | DIPYRIDAMOLE |
| ASPIRIN/CAFFEINE | EPHEDRINE/ASPIRIN/ACETANILIDE/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE | HYDROCODONE BITARTRATE/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM | METHOCARBAMOL/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE | ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE CITRATE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE HCL | OXYCODONE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID | PENTAZOCINE HCL/ASPIRIN |
| ASPIRIN/DIPYRIDAMOLE | PHENYLEPHRINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN |
| ASPIRIN/MEPROBAMATE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE |
| ASPIRIN/SALICYLAMIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE |
| ASPIRIN/SODIUM BICARBONATE/CITRIC ACID | PRASUGREL HCL |
| BUTALBITAL/ASPIRIN/CAFFEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| CARISOPRODOL/ASPIRIN | PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN | TICAGRELOR |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN | V ORAPAXAR SULFATE |
| NDC Brand Name | |
| ARTHRITIS PAIN | BAYER ASPIRIN |
| ARTHRITIS PAIN FORMULA | BAYER ASPIRIN MAXIMUM |
| ARTHRITIS PAIN FORMULA A-F | ECOTRIN |
| ARTHRITIS PAIN RELIEF | ECOTRIN MAXIMUM STRENGTH |
| ARTHRITIS PAIN RELIEVER | MAPAP ARTHRITIS PAIN |
| BAYER ARTHRITIS PAIN REGIMEN | PLAVIX |

## Angiotensin II Receptor Blockers

| NDC Generic Name | |
|---|---|
| ALISKIREN/VALSARTAN | LOSARTAN POTASSIUM |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE |
| AMLODIPINE BESYLATE/VALSARTAN | OLMESARTAN MEDOXOMIL |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZID |
| AZILSARTAN MEDOXOMIL | OLMESARTAN MEDOXOMIL/HYDROCHLOROTHIAZIDE |
| AZILSARTAN MEDOXOMIL/CHLORTHALIDONE | TELMISARTAN |
| CANDESARTAN CILEXETIL | TELMISARTAN/AMLODIPINE BESYLATE |
| CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE | TELMISARTAN/HYDROCHLOROTHIAZIDE |
| IRBESARTAN | VALSARTAN |

| IRBESARTAN/HYDROCHLOROTHIAZIDE | VALSARTAN/HYDROCHLOROTHIAZIDE | |
|--------------------------------|--------------------------------|---|
| NDC Brand Name | | |
| AMLODIPINE-VALSARTAN | EXFORGE HCT | |
| ATACAND | HYZAAR | |
| ATACAND HCT | IRBESARTAN | |
| AVALIDE | IRBESARTAN-HYDROCHLOROTHIAZIDE | |
| AVAPRO | LOSARTAN POTASSIUM | |
| AZOR | LOSARTAN-HYDROCHLOROTHIAZIDE | |
| BENICAR | MICARDIS | |
| BENICAR HCT | MICARDIS HCT | |
| CANDESARTAN CILEXETIL | TELMISARTAN | |
| CANDESARTAN-HYDROCHLOROTHIAZID | TELMISARTAN-AMLODIPINE | |
| COZAAR | TELMISARTAN-HYDROCHLOROTHIAZID | |
| DIOVAN | TRIBENZOR | |
| DIOVAN HCT | TWYNSTA | |
| EDARBI | VALSARTAN | |
| EDARBYCLOR | VALSARTAN-HYDROCHLOROTHIAZIDE | |
| EXFORGE | VALTURNA | · |

| Angiotensin Converting Enzyme inhibitors | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | LISINOPRIL |
| BENAZEPRIL HCL | LISINOPRIL/HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE | MOEXIPRIL HCL |
| CAPTOPRIL | MOEXIPRIL HCL/HYDROCHLOROTHIAZIDE |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | PERINDOPRIL ERBUMINE |
| ENALAPRIL MALEATE | QUINAPRIL HCL |
| ENALAPRIL MALEATE/FELODIPINE | QUINAPRIL HCL/HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE | RAMIPRIL |
| ENALAPRILAT DIHYDRATE | TRANDOLAPRIL |
| FOSINOPRIL SODIUM | TRANDOLAPRIL/VERAPAMIL HCL |
| FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ACCUPRIL | LOTREL |
| ACCURETIC | LYTENSOPRIL |
| ACEON | LYTENSOPRIL-90 |
| ALTACE | MAVIK |
| AMLODIPINE BESYLATE-BENAZEPRIL | MOEXIPRIL HCL |
| BENAZEPRIL HCL | MOEXIPRIL-HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL-HCTZ | MONOPRIL |
| BENAZEPRIL-HYDROCHLOROTHIAZIDE | MONOPRIL HCT |
| CAPOTEN | PERINDOPRIL ERBUMINE |
| CAPOZIDE | PRINIVIL |
| CAPTOPRIL | PRINZIDE |
| CAPTOPRIL-HYDROCHLOROTHIAZIDE | QUINAPRIL |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | QUINAPRIL HCL |
| ENALAPRIL MALEATE | QUINAPRIL-HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE-HCTZ | QUINARETIC |
| ENALAPRIL MALEATE/HCTZ | RAMIPRIL |
| ENALAPRIL-HYDROCHLOROTHIAZIDE | TARKA |
| ENALAPRILAT | TRANDOLAPRIL |
| EPANED | TRANDOLAPRIL-VERAPAMIL |
| FOSINOPRIL SODIUM | UNIRETIC |
| FOSINOPRIL-HYDROCHLOROTHIAZIDE | UNIVASC |
| LEXXEL | VASERETIC |
| LISINOPRIL | VASOTEC |
| LISINOPRIL-HCTZ | VASOTEC I.V. |
| LISINOPRIL-HYDROCHLOROTHIAZIDE | ZESTORETIC |
| LOTENSIN | ZESTRIL |
| LOTENSIN HCT | |

#### Beta blockers

| Deta blockers | |
|-------------------------|------------------------------------------|
| NDC Generic Name | |
| ACEBUTOLOL HCL | ESMOLOL HCL |
| ATENOLOL | LABETALOL HCL |
| ATENOLOL/CHLORTHALIDONE | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE |
| BISOPROLOL FUMARATE | METOPROLOL TARTRATE |

| BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE | METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE |
|---|---|
| BRIMONIDINE TARTRATE/TIMOLOL MALEATE | NEBIVOLOL HCL |
| CARTEOLOL HCL | SOTALOL HCL |
| CARVEDILOL | TIMOLOL |
| CARVEDILOL PHOSPHATE | TIMOLOL MALEATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE | TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE/PF | TIMOLOL MALEATE/PF |
| NDC Brand Name | |
| ACEBUTOLOL HCL | ISTALOL |
| ATENOLOL | KERLONE |
| ATENOLOL W/CHLORTHALIDONE | LABETALOL HCL |
| ATENOLOL-CHLORTHALIDONE | LOPRESSOR |
| BETAPACE | LOPRESSOR HCT |
| BETAPACE AF | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL TARTRATE |
| BETIMOL | METOPROLOL-HYDROCHLOROTHIAZIDE |
| BETOPTIC | NORMODYNE |
| BETOPTIC S | OCUPRESS |
| BISOPROLOL FUMARATE | SECTRAL |
| BISOPROLOL FUMARATE-HCTZ | SENORMIN |
| BISOPROLOL FUMARATE/HCTZ | SORINE |
| BISOPROLOL-HYDROCHLOROTHIAZIDE | SOTALOL |
| BLOCADREN | SOTALOL AF |
| BREVIBLOC | SOTALOL HCL |
| BYSTOLIC | TENORETIC 100 |
| CARTEOLOL HCL | TENORETIC 50 |
| CARTROL | TENORMIN |
| CARVEDILOL | TENORMIN CALENDAR PAK |
| COMBIGAN | TIMOLIDE |
| COREG | TIMOLOL MALEATE |
| COREG CR | TIMOPTIC |
| COSOPT | TIMOPTIC OCUDOSE |
| COSOPT PF | TIMOPTIC-XE |
| DORZOLAMIDE-TIMOLOL | TOPROL XL |
| DUTOPROL | TRANDATE |
| ESMOLOL HCL | ZEBETA |
| HYPERTENSOLOL | ZIAC |

#### Calcium channel blockers

| Calcium channel blockers | |
|---|---|
| HCPCS | |
| C9248 | |
| NDC Generic Name | |
| ALISKIREN HEMIFUMARATE/AMLODIPINE BESYLATE | BEPRIDIL HCL |
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE | CLEVIDIPINE BUTYRATE |
| AMLODIPINE BESYLATE | DILTIAZEM HCL |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | DILTIAZEM HCL/DEXTROSE 5 % IN WATER |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | DILTIAZEM MALATE |
| AMLODIPINE BESYLATE/VALSARTAN | ENALAPRIL MALEATE/FELODIPINE |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ADALAT | ISOPTIN |
| ADALAT CC | ISOPTIN SR |
| AFEDITAB CR | ISRADIPINE |
| AMLODIPINE BESILATE | LEXXEL |
| AMLODIPINE BESYLATE | LOTREL |
| AMLODIPINE BESYLATE-BENAZEPRIL | MATZIM LA |
| AMLODIPINE-ATORVASTATIN | NICARDIPINE HCL |
| AMLODIPINE-VALSARTAN | NICARDIPINE HCL-D5W |
| AMTURNIDE | NIFEDIAC CC |
| AZOR | NIFEDICAL XL |
| CADUET | NIFEDIPINE |
| CALAN | NIFEDIPINE ER |
| CALAN SR | NIFEDIPINE XL |
| CARDENE | NIMODIPINE |
| CARDENE I.V. | NIMOTOP |
| CARDENE SR | NISOLDIPINE |
| CARDIZEM | NORVASC |

| NYMALIZE |
|------------------------|
| PLENDIL |
| POSICOR |
| PROCARDIA |
| PROCARDIA XL |
| SULAR |
| TARKA |
| TAZTIA XT |
| TEKAMLO |
| TELMISARTAN-AMLODIPINE |
| TIAMATE |
| TIAZAC |
| TRANDOLAPRIL-VERAPAMIL |
| TRIBENZOR |
| TWYNSTA |
| VASCOR |
| VERAPAMIL ER |
| VERAPAMIL ER PM |
| VERAPAMIL HCL |
| VERAPAMIL SR |
| VERELAN |
| VERELAN PM |

#### Diuretics

| NDC Generic Name | |
|-----------------------------------|---------------------|
| AMILORIDE HCL | HYDROCHLOROTHIAZIDE |
| AMILORIDE HCL/HYDROCHLOROTHIAZIDE | HYDROFLUMETHIAZIDE |
| BENDROFLUMETHIAZIDE | INDAPAMIDE |
| BUMETANIDE | METHYCLOTHIAZIDE |
| CHLOROTHIAZIDE | METOLAZONE |
| CHLORTHALIDONE | POLYTHIAZIDE |
| EPLERENONE | SPIRONOLACTONE |
| ETHACRYNATE SODIUM | TORSEMIDE |
| ETHACRYNIC ACID | TRIAMTERENE |
| FUROSEMIDE | TRICHLORMETHIAZIDE |

## Nitrates

| Nitrates | |
|---|---|
| NDC Generic Name | |
| ISOSORBIDE DINITRATE | NITROGLYCERIN |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL | NITROGLYCERIN/DEXTROSE 5 % IN WATER |
| ISOSORBIDE MONONITRATE | RANOLAZINE |
| NDC Brand Name | |
| ANG-O-SPAN | NITRO-TRANS SYSTEM |
| ANGINABID | NITRO-TRANSDERMAL |
| BIDIL | NITRO-TRANSDERMAL SYSTEM |
| CARDABID | NITROBART |
| DEPONIT | NITROCAP |
| DILATRATE-SR | NITROCINE |
| IMDUR | NITROCOT |
| ISD | NITRODISC |
| ISMO | NITROGARD |
| ISO-BID | NITROGLYCERIN |
| ISO-D | NITROGLYCERIN IN D5W |
| ISOCHRON | NITROGLYCERIN PATCH |
| ISODITRATE | NITROGLYCERIN T/R |
| ISONATE | NITROGLYN |
| ISONATE TR | NITROGYLCERIN |
| ISOR-BID | NITROL |
| ISORDIL | NITROLINGUAL |
| ISORDIL TITRADOSE | NITROMED |
| ISOREX-10 | NITROMIST |
| ISOREX-2.5 | NITRONAL |
| ISOREX-5 | NITRONG |
| ISOSORBIDE DINITRATE | NITROQUICK |
| ISOSORBIDE MONONITRATE | NITROREX |
| ISOSORBIDE MONONITRATE ER | NITROSPAN |
| ISOTRATE | NITROSTAT |

| ISOTRATE ER | NITROSTAT IV |
|--------------------------|-----------------|
| KENSORBIDE | NITROSTAT SR |
| LEMOTRATE | NITROTAB |
| MI-TRATES 2.5 | NITROTYM |
| MI-TRATES 6.5 | NTG |
| MINITRAN | NTS |
| MONOKET | ONSET-10 |
| N-G-C | ONSET-5 |
| N.T.S. | RANEXA |
| NITREK | RECTIV |
| NITRO | SORATE-2.5 |
| NITRO MAST TIMED RELEASE | SORATE-40 |
| NITRO S.A. | SORATE-5 |
| NITRO T.D. | SORBATE-10 |
| NITRO TRANSDERM | SORBATE-5 |
| NITRO TRANSDERMAL | SORBIDE |
| NITRO-BID | SORBITRATE |
| NITRO-BID IV | SORBITRATE SA |
| NITRO-CAPS TIME DOSE | TRANSDERM-NITRO |
| NITRO-DUR | TRATES |
| NITRO-PAR | TRIDIL |
| NITRO-TD-ACA | WF-NITRO |
| NITRO-TIME | |

Lipid lowering drugs

| Lipid lowering drugs | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | METHYLTETRAHYDROFOLATE GLUCOSAMINE/NIACINAMIDE/CUPRIC &ZN OX |
| ARGININE/NIACIN/YOHIMBE BARK/GINSENG/GNK/DAMIANA/SCHISANDRA | NIACIN |
| ATORVASTATIN CALCIUM | NIACIN (INOSITOL NIACINATE) |
| BETA-CAROTENE(A) W-C & E/NIACINAMIDE/VIT B2/LUT/MIN/GLU-ONE | NIACIN/CAPSAICIN/YOHIMBE BARK/GINSENG/GNK BI EX/DAMIANA/OATS |
| CERAMIDES 1,3,6-11/NIACINAMIDE | NIACIN/LOVASTATIN |
| CERAMIDES 1,3,6-11/NIACINAMIDE/HYALURONIC ACID | NIACIN/SIMVASTATIN |
| CHOLESTYRAMINE | NIACINAMIDE |
| CHOLESTYRAMINE (WITH SUGAR) | NIACINAMIDE ASCORBATE |
| CHOLESTYRAMINE/ASPARTAME | NIACINAMIDE/AZELAIC ACID/ZINC OXIDE/VIT B6/COPPER/FA |
| COLESEVELAM HCL | NIACINAMIDE/RIBOFLAVIN/BETA-CAROTENE(A) W-C & E/MINERALS |
| COLESTIPOL HCL | NIACINAMIDE/VIT B6/VIT C/FA/COPPER/MG CIT/ZN GLUC/ALIP ACID |
| EZETIMIBE | PECTIN/INOSITOL/BIOFLAVONOIDS/NIACIN/SOYBEAN |
| EZETIMIBE/ATORVASTATIN CALCIUM | PITAVASTATIN CALCIUM |
| EZETIMIBE/SIMVASTATIN | POLICOSANOL/INOSITOL NIACINATE/GARLIC |
| FENOFIBRATE | PRAVASTATIN SODIUM |
| FENOFIBRATE NANOCRYSTALLIZED | ROSUVASTATIN CALCIUM |
| FENOFIBRATE, MICRONIZED | SIMVASTATIN |
| FLUVASTATIN SODIUM | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| FOLIC ACID/NIACINAMIDE/CUPRIC OXIDE/ZINC OXIDE | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/CYANOCOBALAMIN/PROTEASE |
| FOLIC ACID/NIACINAMIDE/ZINC | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/DEXPANTHENOL/PYRIDOXINE |
| GEMFIBROZIL | THIAMINE M.NIT/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/C/FA |
| INOSITOL NIACINATE | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/VIT C/FA |
| IRON FUMARATE & POLYSAC COMP/FOLIC ACID/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
| IRON FUMARATE & POLYSAC COMP/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL | VIT B2/NIACINAMIDE/PYRIDOXINE HCL/CYANOCOBALAMIN/D-PANTHENOL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN | VIT C/PYRIDOXINE HCL/NIACIN/FA/VIT B12/HERBAL COMPLEX NO.192 |
| LOVASTATIN | VITAMIN B COMPLEX NO.12/NIACINAMIDE |
| LYSINE HCL/NIACINAMIDE/THIAMINE | VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 | |

#### Non-insulin diabetes medications

| Non-insulin diabetes inedications | |
|--------------------------------------|-------------------------------------|
| NDC Generic Name | |
| ACARBOSE | MIGLITOL |
| ACETOHEXAMIDE | NATEGLINIDE |
| ALOGLIPTIN BENZOATE | PIOGLITAZONE HCL |
| ALOGLIPTIN BENZOATE/METFORMIN HCL | PIOGLITAZONE HCL/GLIMEPIRIDE |
| ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL | PIOGLITAZONE HCL/METFORMIN HCL |
| CANAGLIFLOZIN/METFORMIN HCL | REPAGLINIDE |
| CHLORPROPAMIDE | REPAGLINIDE/METFORMIN HCL |
| GLIMEPIRIDE | ROSIGLITAZONE MALEATE |
| GLIPIZIDE | ROSIGLITAZONE MALEATE/GLIMEPIRIDE |
| GLIPIZIDE/METFORMIN HCL | ROSIGLITAZONE MALEATE/METFORMIN HCL |

| GLYBURIDE | SAXAGLIPTIN HCL |
|---|---|
| GLYBURIDE/METFORMIN HCL | SAXAGLIPTIN HCL/METFORMIN HCL |
| LINAGLIPTIN | SITAGLIPTIN PHOSPHATE |
| LINAGLIPTIN/METFORMIN HCL | SITAGLIPTIN PHOSPHATE/METFORMIN HCL |
| METFORMIN HCL | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE | TOLAZAMIDE |
| METFORMIN/CAFFEINE/AMINO ACIDS#7/HERBAL COMB#125/CHOLINE BIT | TOLBUTAMIDE |
| NDC Brand Name | |
| ACARBOSE | ICN-TOLAM |
| ACETOHEXAMIDE | INSULASE |
| ACTOPLUS MET | INVOKAMET |
| ACTOPLUS MET XR | JANUMET |
| ACTOS | JANUMET XR |
| AMARYL | JANUVIA |
| APPFORMIN | JENTADUETO |
| APPFORMIN-D | JUVISYNC |
| AVANDAMET | KAZANO |
| AVANDARYL | KOMBIGLYZE XR |
| AVANDIA | METAGLIP |
| CHLORABETIC 250 | METFORMIN HCL |
| CHLORPROPAMIDE | METFORMIN HCL ER |
| DIABETA | MICRONASE |
| DIABINESE | NATEGLINIDE |
| DIBATROL | NESINA |
| DUETACT | ONGLYZA |
| DYMELOR | ORIBETIC |
| FORTAMET | ORINASE |
| GLIMEPIRIDE | OSENI |
| GLIPIZIDE | PIOGLITAZONE HCL |
| GLIPIZIDE ER | PIOGLITAZONE-GLIMEPIRIDE |
| GLIPIZIDE XL | PIOGLITAZONE-METFORMIN |
| GLIPIZIDE-METFORMIN | PRANDIMET |
| GLUCAMIDE | PRANDIN |
| GLUCOPHAGE | PRECOSE |
| GLUCOPHAGE XR | REPAGLINIDE |
| GLUCOTROL | RIOMET |
| GLUCOTROL XL | RONASE |
| GLUCOVANCE | SK-TOLBUTAMIDE |
| GLUMETZA | STARLIX |
| GLYBURIDE | TOLAMIDE |
| GLYBURIDE MICRONIZED | TOLAZAMIDE |
| GLYBURIDE-METFORMIN HCL | TOLBUTAMIDE |
| GLYCRON | TOLINASE |
| GLYNASE | TRADJENTA |
| GLYSET | |

## Insulin


| EXUBERA COMBINATION PACK 12 | INSULIN NPH BEEF |
|-----------------------------|--------------------------------|
| EXUBERA COMBINATION PACK 15 | INSULIN NPH PURIFIED PORK |
| EXUBERA KIT | INSULIN R PORK PURIFIED |
| EXUBERA PATIENT PACK | INSULIN R PURIFIED PORK |
| HUMALOG | INSULIN REGULAR PORK |
| HUMALOG MIX 50-50 | INSULIN REGULAR PURIFIED PORK |
| HUMALOG MIX 50/50 | ISOPHANE INSULIN BEEF |
| HUMALOG MIX 75-25 | ISOPHANE PURIFIED BEEF INSULIN |
| HUMULIN 50-50 | LANTUS |
| HUMULIN 70-30 | LANTUS SOLOSTAR |
| HUMULIN 70/30 | LENTE INSULIN BEEF |
| HUMULIN 70/30 KWIKPEN | LEVEMIR |
| HUMULIN BR | LEVEMIR FLEXPEN |
| HUMULIN L | LEVEMIR FLEXTOUCH |
| HUMULIN N | MONOTARD HUMAN LENTE |
| HUMULIN N KWIKPEN | NOVOLIN 70-30 |
| HUMULIN R | NOVOLIN 70-30 INNOLET |
| HUMULIN U | NOVOLIN 70/30 |
| ILETIN I LENTE | NOVOLIN L |
| ILETIN I NPH | NOVOLIN N |
| ILETIN I REGULAR | NOVOLIN N INNOLET |
| ILETIN I SEMILENTE | NOVOLIN R |
| ILETIN I ULTRALENTE | NOVOLOG |
| ILETIN II LENTE(BEEF) | NOVOLOG FLEXPEN |
| ILETIN II LENTE(PORK) | NOVOLOG MIX 70-30 |
| ILETIN II NPH(BEEF) | NOVOLOG MIX 70-30 FLEXPEN |
| ILETIN II NPH(PORK) | PROTAMINE ZINC INSULIN BEEF |
| ILETIN II REGULAR(BEEF) | PURIFIED BEEF INSULIN ZINC |
| ILETIN II REGULAR(PORK) | PURIFIED PORK INSULIN |
| ILETIN II REGULAR(PORK)CONC | VELOSULIN HUMAN |
| INSULATARD HUMAN N | VELOSULIN HUMAN BR |
| INSULATARD N | VELOSULIN HUMAN R |
| INSULATARD NPH HUMAN | VELOSULIN R |
| INSULIN L PURIFIED PORK | ZINC |
| INSULIN LENTE BEEF | |

#### Antidepressants

| HCPCS | |
|---|---|
| J1320 | |
| NDC Generic Name | |
| AMITRIPTYLINE HCL | IMIPRAMINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE PAMOATE |
| AMOXAPINE | ISOCARBOXAZID |
| BUPROPION HBR | LEVOMILNACIPRAN HYDROCHLORIDE |
| BUPROPION HCL | MAPROTILINE HCL |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB15 | MIRTAZAPINE |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB16 | NEFAZODONE HCL |
| CITALOPRAM HYDROBROMIDE | NORTRIPTYLINE HCL |
| CLOMIPRAMINE HCL | OLANZAPINE/FLUOXETINE HCL |
| DESIPRAMINE HCL | PAROXETINE HCL |
| DESVENLAFAXINE | PAROXETINE MESYLATE |
| DESVENLAFAXINE FUMARATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| DESVENLAFAXINE SUCCINATE | PHENELZINE SULFATE |
| DOXEPIN HCL | PROTRIPTYLINE HCL |
| DULOXETINE HCL | SERTRALINE HCL |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| FLUOXETINE | TRAZODONE HCL/DIETARY SUPPLEMENT, MISC. COMBO8 |
| FLUOXETINE HCL | TRIMIPRAMINE MALEATE |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC COMB17 | VENLAFAXINE HCL |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 | VILAZODONE HYDROCHLORIDE |
| FLUVOXAMINE MALEATE | VORTIOXETINE HYDROBROMIDE |
| NDC Brand Name | |
| ADAPIN | LIMBITROL DS |
| AMITID | LUDIOMIL |
| AMITRIPTYLINE HCL | LUVOX |
| AMITRIPTYLINE W/PERPHENAZINE | LUVOX CR |
| AMITRIPTYLINE-CHLORDIAZEPOXIDE | MAPROTILINE HCL |
| AMITRIPTYLINE-PERPHENAZINE | MARPLAN |

| AMONAPINE MINTAZAPHE ANYDROUS ANAPETAMIN PREDITAMONE PREDITAMONE NOFERAMIN NEFACOONE HCI NOFERAMIN NEFACOONE HCI NOFERAMIN NOFERAMIN NOFERAMIN NOFERAMIN NORTRIPTYLIN HCI OLANZARIMA HCI OLANZARIMA HCI SENDERIMA SENDER PAMELOR BUDEPRION SR BUDEPRION SR BUDEPRION SR PAMELOR BUDEPRION SR PARIC CR BUDEPRION MCI PARIC CR BUDEPRION MCI PARIC CR BUDEPRION MCI PERTIND BUDEPRION HCI PERTIND PERTIND BUDEPRION HCI PERTIND BUDEPRION HCI PERTIND BUDEPRION HCI PERTIND PERTIND BUDEPRION HCI BUDEPRION HCI PERTIND BUDEPRION HCI BUDE | AMITRIPTYLINE/CHLORDIAZEPOXIDE | MIRTAZAPINE |
|---|---|---|
| AMAFABIL APRIEZIM NARONE APPRITAMONE NOBERAMI NO | · | |
| NEFACOONE INC. | | |
| MORFRANII | | |
| APSENDIN MORTAMINE HU. APSENDIN MORTAMINE HU. AVENITY HU. BRIDDERICO MORTAMINE HU. AVENITY HU. BRIDDERICO MORTAMINE HU. AVENITY HU. BRIDDERICO M. BR | | |
| ASENDIN | | |
| AVENTYL HCL OLANAZARIK-FLUXXETINE HCL BRISTELIX BRISTELIX BRISTELIX DEFPROR N. BRISTELIX PARKICR BLUDEPRON X. PEXEVA PEXEVA PEXEVA PROSE BLUPROPHON X. BLUPROPHON X. BLUPROPHON X. PEXEVA PROSE BLUPROPHON X. BLUPROPHON X. PROSE BLUPROPHON X. PROSE BLUPROPHON X. BLUDEPROPHON X. PROSE BLUPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUD X. BLUDEPROPHON X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDR | | |
| SINTELLIX OLEFTO & R | | |
| RRISDELLE PAMELOR PARCETINE H.C. PERPERBAN PARCETINE H.C. PERPERBAN PERPENBAN PERPENBA | | |
| BRUDEPRION SR | | |
| PAXIL PAXI | | |
| BURDEDAN PAXIL CR | | |
| BURDOPION H.C. PERTER | | |
| BURDOPION HCL ER BURDOPION HCL SR BURDOPION SC PEXEVA BURDOPION SC PEXEVA BURDOPION SC PERCENA PRISTIQ ER BURDOPION SC PROTECT | | |
| BURDOPION HCL SR | | |
| PURPOPION XL | | |
| CELEXA PROTREPTYLINE HCL CHTALOPRAM PROZAC CITALOPRAM HRR PROZAC REHIVE DESIPRAM DESVENLA FAXINE FULL SERTRON DESVENLA FAXINE FULL SERTRON SELFEMRA DULOXETINE HCL SERTRALINE HCL TRAVIL 10-2 | | |
| CHIORDIAZEPOXIDE-AMITRIPTYUNE PROZAC CITALOPRAM PROZAC CWERKLY PRUDOXIN CYMBALTA Q.E. L DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RE-LUVE DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FUMARATE ER SARAFEM SELFEMRA DOKERIH HCL SENTROXATINE DOLOXETINE HCL SERTROXATINE DOLOXETINE HCL SERTROXATINE DOLOXETINE HCL SERTROXATINE PROLOXE PVILL 10 SERZONE PVILL 25 SINEQUAN SK-PAMITRIPTYUNE SK-PAMITRIPTY | | |
| CITALOPRAM HBR PROZAC C TITALOPRAM HBR PROZAC WEEKLY CICMIPPAMINE HCL PRUDOWN CYMBALTA Q.E.L PRUDOWN CICMIPPAMINE HCL PRUDOWN CESTINAL Q.E.L PRUDOWN DESIPHARMINE HCL RAPPILUX DESIPHARMINE HCL REHVE DESIPHARMINE HCL REHVE DESIVENLARAKINE ER REMERON DESVENLARAKINE ER SARAFEM DESVENLARAKINE FUMARATE ER SARAFEM DOXEPIN HCL SENTROXATINE DULOXEINIE HCL SERTRALINE SERTRALINE SER | | |
| PROZAC WEEKLY | | |
| PRIDOXIN | | |
| CYMBALTA | | |
| DECONIL RAPIFLUX DESSIPRAMINE HCL RE-UVE DESSIPRAMINE HCL RE-UVE REMERON DESSIPRAMINE FUNARATE ER REMERON DESSURLAFAXINE FUMARATE ER SELFEMRA DOXEDIH HCL SERTROWATINE DOULOXETINE HCL SERTROWATINE SELFEMRA SILENOR E-VILL 100 SILENOR E-VILL 100 SILENOR E-VILL 55 SINEQUAN SERVALISO SK-AMITIRIPTYLINE E-VILL 50 SK-AMITIRIPTYLINE E-VILL 75 SK-PAMINE STABANIL STEFEXOR STABANIL SURMONTIL E-FEXOR SURMONTIL E-BAYL SURMONTIL E-MITRIP TOFRANIL-PM FINOVIL SYMBYAX SURMONTIL E-MITRIP TOFRANIL-PM FINOVIL TRAZAMINE E-SOTTALOPRAM OXALATE TRAZODONE HCL E-TRAFON 2-10 TRIAVIL 1-0 E-TRAFON 2-10 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-10 TRIAVIL 1-10 | | |
| DESIPRAMINE HCL DESVENLAFAXINE FUMARATE ER DESVENLAFAXINE MCL DULOXETINE HCL SERTROLATINE SERTROLATINE SERTROLATION SERTROLATINE SERTROLATION | | · · |
| DESVENLAFAXINE ER DESVENLAFAXINE FUMARATE ER DESYREL SELFEMRA DOXEPIN HCL SENTROXATINE DULOXETINE HCL SERTRALINE HCL SILENOR SILENOR SILENOR SILENOR SERTRALINE SIMEQUAN SERTRALINE SERTRALINE SERTRALINE SERTRALINE SERTRALINE SERTRALINE SERTRALINE SOUTH TOFARAIL FINAPIL ENOPTH ENOPTH SERTRALINE SECTIALOPRAM OXALATE TRAZODONE HCL TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-5 TRANIL 2-6 TRANIL 2-7 TRANIL 2-7 TRANIL 2-8 TRANIL 2-9 TRANIL 2-9 TRANIL 2-10 TRANIL 2-1 | | |
| DESVENLAFAXINE FUMARATE ER DESVERL DESVERL DESVERL SELFEMRA DOUCKPIN HCL SENTROXATINE DULOXETINE HCL SERTALINE HCL SE | | |
| DESYREL DESYREL DESYREL DESPIRACATINE DOXEPIN HCL SENTROXATINE DUICNETINE HCL SENTROXATINE DUICNETINE HCL SERZONE E-VILL 100 SIRNOR E-VILL 25 SINEQUAN SEVILL 25 SINEQUAN SK-RAMITRIPTYLINE E-VILL 50 SK-RAMITRIPTYLINE E-VILL 57 SK-PRAMINE STABANIL STABANIL STABANIL STABANIL SEFEXOR STABANIL SEMMONTIL ELAVIL SYMBYAX EMITRIP TOFRANIL FINDEP TOFRANILPM FINOVIL TRAZAMINE SECTIALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRAVIL 2-10 ETRAFON 2-10 TRAVIL 2-10 ETRAFON 2-10 TRAVIL 2-10 ETRAFON 4-10 TRAVIL 2-10 ETRAFON 4-10 TRAVIL 2-10 ETRAFON A-10 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON TORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-20 ETRAFON BORTE 4-25 TRAVIL 2-3 ETRAFON BORTE 4-25 TRAVIL 2-3 ETRAFON BORTE 4-25 TRAVIL 2-3 ETRAFON BORTE 4-3 TRAVIL 2-10 TRAVIL 2-10 TRAVIL 2-10 TRAVIL 2-10 TRAVIL 2-10 TRAVIL 2-10 TRAVIL 2-10 TRA | | |
| DOUCRPIN HCL SERTRALINE HCL SILENOR SILENOR SILENOR SILENOR SILENOR SEAMITRIPTYLINE EVILL 75 SEPRAMINE SEFEXOR STABANIL SEFEXOR STABANIL SUMMONTIL SELAVIL SYMBYAX SILENOR SILENOR STABANIL SYMBYAX SILENOR STABANIL SELAVIL SELAVIL SELAV | | |
| DULOXETINE HCL SERTABLINE HCL SERZONE E-VILL 10 SERZONE E-VILL 25 SINEQUAN SILENOR E-VILL 25 SINEQUAN SINEQUAN SEPERSOR SEPERSOR STABANIL SEFEXOR STABANIL EFFEXOR STABANIL EFFEXOR SYMBYAX SUMMONTIL LAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRIAVIL 2-10 TETRAFON 2-25 TRIAVIL 2-25 ETRAFON 2-10 TRIAVIL 2-25 ETRAFON 4-10 TRIAVIL 2-25 ETRAFON 1-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-30 TRIAVIL 2-4 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-6 ETRAFON FORTE 4-25 TRIAVIL 2-7 TRIAVIL 2-8 ETRAFON FORTE 4-25 TRIAVIL 2-9 ETRAFON FORTE 4-25 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-26 ETRAFON FORTE 4-25 TRIAVIL 2-30 TRIAVIL 2-4 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-10 TRIAVI | | |
| E-VILL 10 SERZONE E-VILL 100 SILENOR E-VILL 25 SINEQUAN E-VILL 50 SK-AMITRIPTYLINE E-VILL 75 SK-PRAMINE EFFEKOR STABANIL EFFEKOR STABANIL EFFEKOR XR SURMONTIL LAVIL SYMBYAX EMITIRP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNAFOR 2-10 TRIAVIL 2-10 ETRAFON 3-10 TRIAVIL 2-10 ETRAFON 3-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 1-10 TRIAVIL 2-10 | | |
| E-VILL 25 SINEQUAN E-VILL 25 SINEQUAN E-VILL 25 SINEQUAN E-VILL 75 SK-PRAMINE EFFEXOR STABANIL EFFEXOR STABANIL EFFEXOR STABANIL ELAVIL SYMBYAX EMITRIP ELAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENCOPLE ENCOPL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-10 ETRAFON 6-10 ETRAFON FORTE 4-25 ETRAFON FORTE 4-25 ETRAFON FORTE 4-25 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-5 FETRAFON FORTE 4-25 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-5 FETRAFON TRIAVIL 5- | | |
| SINEQUAN | | |
| E-VILL 50 E-VILL 75 SK-PRAMINE EFFEXOR STABANIL EFFEXOR STABANIL EFFEXOR SYMBYAX ELAVIL SYMBYAX ELAVIL ELAVIL SYMBYAX ENTIFIP TOFRANIL-PM ENOUTH ENOUTH ENOUTH ENOUTH ENOUTH ETRACODONE HCL ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON BORTH 4-25 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2 | | |
| SK-PRAMINE | | |
| EFFEXOR STABANIL EFFEXOR XR SURMONTIL ELAVIL SYMBYAX EMITRP TOFRANIL ENDEP TOFRANIL-PM ENOVIL TRAZAMINE ENOVIL TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-5 ETRAFON 2-25 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 EFETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-10 FLUOX | | |
| SURMONTIL | | |
| ELAVIL SYMBYAX | | |
| EMITRIP ENDEP TOFRANIL ENDEP TOFRANILPM ENOVIL ENOVIL ENOVIL ETRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 TRIAVIL 2-5-2 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-50 FLUOVAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLOVOXAMINE MALEATE FLOVATE FORFIVO XL SABOXETINE VENLAFAXINE HCL MINAVATE | | |
| ENDEP FINDER FIN | | STIVIDIAX |
| ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUOXEMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIMIPRAMINE MALEATE TRIMIPRAMINE MALEATE TRIMIPRAMINE HCL TRIAVIL 4-50 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 2-25 TRIAVIL | I E M I T D D | TOFRANII |
| TRAZODONE HCL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-6 FETZIMA TRIAVIL 2-7 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FORFIVO XL GABOXETINE GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL ER WANATE MIPPRAMINE HCL WINACTIL MIPRAMINE PAMOATE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 4-10 TRIAVIL 2-5 TRIAVIL 2-10 TRIAVIL 2-1 | EMITRIP | |
| ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 25-2 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FURD YENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL WENLAFAXINE HCL ER WANATE WIBRYD WIBRYD WIBRYD WIBRYD WIBRYD WIBRYD WIBRYD WINFRAMINE HCL WINFRAMINE HCL WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT ZONALON | ENDEP | TOFRANIL-PM |
| ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FULOXETINE DR TRIAVIL 4-25 FULOXETINE HCL TRIAVIL 4-50 FULVOXAMINE MALEATE TRIMIPRAMINE MALEATE FULVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER IMIPRAMINE HCL VIVACTIL IMIPRAMINE HCL VIVACTIL IMIPRAMINE PAMOATE WELBUTRIN JANIMINE WELBUTRIN SR KENVIL WELBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP<br>ENOVIL | TOFRANIL-PM<br>TRAZAMINE |
| TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR FLUOXETINE HCL TRIAVIL 4-50 FLUOXEMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMIPRAMINE MALEATE FORFIVO XL VENLAFAXINE HCL VENLAFAXINE HCL MIPPAMINE HCL WIBRYD MIPPAMINE HCL WIBRYD WIBRYD MIPPAMINE HCL WINACTIL MIPPAMINE PAMOATE VELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL | ENDEP ENOVIL ESCITALOPRAM OXALATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL |
| TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMPRAMINE MALEATE TRIMPRAMINE MALEATE FORFIVO XL GABOXETINE WENLAFAXINE HCL WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WELBUTRIN JANIMINE JANIMINE KENVIL KHEDEZLA ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 |
| TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE HCL FLUVOXAMINE H | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 |
| TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMIPRAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIBRYD VIBRYD VIMIPRAMINE HCL VIVACTIL VIVACTIL VIMIPRAMINE PAMOATE VELLBUTRIN VELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 |
| TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIBRYD VIMIPRAMINE HCL VIVACTIL VIVACTIL VIMIPRAMINE PAMOATE VELLBUTRIN VELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 |
| FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE WENLAFAXINE HCL VENLAFAXINE HCL ER WIBRYD WIBRYD WIBRYD WIBRYD WIMIPRAMINE HCL WINACTIL WIMIPRAMINE PAMOATE WELLBUTRIN JANIMINE KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 |
| TRIMIPRAMINE MALEATE FLUVOXAMINE MALEATE ER FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIIBRYD VIIBRYD VIIBRYD VIIBRYD VIVACTIL | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 |
| FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIVACTIL MIPRAMINE HCL VIVACTIL MIPRAMINE PAMOATE VELBUTRIN VELBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 |
| FORFIVO XL GABOXETINE WENLAFAXINE HCL ER WAVATE WIBRYD WIFRAMINE HCL WIFRAMINE HCL WIFRAMINE PAMOATE WELLBUTRIN WELLBUTRIN SR KENVIL KHEDEZLA KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 |
| GABOXETINE VENLAFAXINE HCL ER VIIBRYD IMIPRAMINE HCL VIVACTIL IMIPRAMINE PAMOATE WELLBUTRIN IANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO VONLAFAXINE HCL ER VIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE |
| MAVATE VIBRYD MIPRAMINE HCL VIVACTIL MIPRAMINE PAMOATE WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO VIBRYD VIVACTIL VEILBUTRIN SR WELLBUTRIN SL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP |
| MIPRAMINE HCL MIPRAMINE PAMOATE MELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO VIVACTIL WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL |
| IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA LEXAPRO WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER |
| JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD |
| KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL |
| KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN |
| LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |
| | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL |
| LIMBITROL ZYBAN | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT |
| | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA LEXAPRO | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON |

## Appendix A Comorbid conditions

**Atrial Fibrillation** 


| Heart | Fai | Iure |
|-------|-----|------|


Stroke or TIA


| 163312 |
|---|
| cerebral arteries 163319 |
| I63319 |
| I63321 |
| 163322 |
| 163323 43401 Cerebral infarction due to thrombosis of bilateral anterior arteries 163329 43401 Cerebral infarction due to thrombosis of unspecified anterior cerebral thrombosis with cerebral infarction cerebral artery 163331 43401 Cerebral infarction due to thrombosis of right posterior cerebral thrombosis with cerebral infarction cerebral artery |
| 163329 43401 Cerebral infarction due to thrombosis of unspecified anterior cerebral thrombosis with cerebral infarction cerebral artery 163331 43401 Cerebral infarction due to thrombosis of right posterior cerebral thrombosis with cerebral infarction cerebral artery |
| I63331 43401 Cerebral infarction due to thrombosis of right posterior Cerebral thrombosis with cerebral infarction cerebral artery |
| l63332 43401 Cerebral infarction due to thrombosis of left posterior Cerebral thrombosis with cerebral infarction |
| cerebral artery |
| I63333 43401 Cerebral infarction to thrombosis of bilateral posterior Cerebral thrombosis with cerebral infarction arteries |
| 163339 43401 Cerebral infarction due to thrombosis of unspecified posterior Cerebral thrombosis with cerebral infarction cerebral artery |
| I63341 43401 Cerebral infarction due to thrombosis of right cerebellar Cerebral thrombosis with cerebral infarction artery |
| I63342 43401 Cerebral infarction due to thrombosis of left cerebellar Cerebral thrombosis with cerebral infarction artery |
| 163343 43401 Cerebral infarction to thrombosis of bilateral cerebellar Cerebral thrombosis with cerebral infarction arteries |
| 163349 43401 Cerebral infarction due to thrombosis of unspecified Cerebral thrombosis with cerebral infarction cerebellar artery |
| 16339 43401 Cerebral infarction due to thrombosis of other cerebral Cerebral thrombosis with cerebral infarction |
| l636 43401 Cerebral infarction due to cerebral venous thrombosis, Cerebral thrombosis with cerebral infarction |
| nonpyogenic 16340 43411 Cerebral infarction due to embolism of unspecified cerebral Cerebral embolism with cerebral infarction |
| l63411 43411 Cerebral infarction due to embolism of right middle cerebral Cerebral embolism with cerebral infarction |
| l63412 43411 Cerebral infarction due to embolism of left middle cerebral Cerebral embolism with cerebral infarction |
| 163413 43411 Cerebral infarction due to embolism of bilateral middle Cerebral embolism with cerebral infarction |
| cerebral arteries |
| cerebral artery 162421 |
| 163421 43411 Cerebral infarction due to embolism of right anterior Cerebral embolism with cerebral infarction cerebral artery |
| 163422 43411 Cerebral infarction due to embolism of left anterior cerebral Cerebral embolism with cerebral infarction artery |
| 163423 43411 Cerebral infarction due to embolism of bilateral anterior Cerebral embolism with cerebral infarction cerebral arteries |
| 163429 43411 Cerebral infarction due to embolism of unspecified anterior cerebral embolism with cerebral infarction |
| 163431 43411 Cerebral infarction due to embolism of right posterior Cerebral embolism with cerebral infarction cerebral artery |
| I63432 43411 Cerebral infarction due to embolism of left posterior cerebral Cerebral embolism with cerebral infarction |
| artery 163433 43411 Cerebral infarction due to embolism of bilateral posterior Cerebral embolism with cerebral infarction |
| cerebral arteries 163439 43411 Cerebral infarction due to embolism of unspecified posterior Cerebral embolism with cerebral infarction |
| cerebral artery |
| artery artery |


Peripheral vascular disease


| Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right leg with ulceration of thigh 170732 Atherosclerosis of other type of bypass graft(s) of the right leg with ulceration of calf |
|---|
| I70728 |
| extremities with rest pain, other extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the right leg with ulceration of thigh Atherosclerosis of other type of bypass graft(s) of the right |
| I70729 |
| extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right leg with ulceration of thigh 170732 Atherosclerosis of other type of bypass graft(s) of the right |
| I70731 Atherosclerosis of other type of bypass graft(s) of the right leg with ulceration of thigh I70732 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of thigh 170732 Atherosclerosis of other type of bypass graft(s) of the right |
| 170732 Atherosclerosis of other type of bypass graft(s) of the right |
| 170733 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of ankle |
| 170734 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of heel and midfoot |
| 170735 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of other part of foot |
| 170738 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of other part of lower leg |
| 170739 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of unspecified site |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of thigh |
| 170742 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of calf |
| 170743 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of ankle |
| I70744 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of heel and midfoot |
| 170745 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of other part of foot |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of other part of lower leg |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of unspecified site |
| Atherosclerosis of other type of bypass graft(s) of other |
| extremity with ulceration |
| Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, right leg |
| Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, left leg 170763 Atherosclerosis of other type of bypass graft(s) of the |
| I70763 Atherosclerosis of other type of bypass graft(s) of the extremities with gangrene, bilateral legs |
| 170768 Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, other extremity |
| 170769 Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, unspecified extremity |
| 170791 Other atherosclerosis of other type of bypass graft(s) of the |
| extremities, right leg |
| 170792 Other atherosclerosis of other type of bypass graft(s) of the |
| extremities, left leg |
| 170793 Other atherosclerosis of other type of bypass graft(s) of the |
| extremities, bilateral legs |
| 170798 Other atherosclerosis of other type of bypass graft(s) of the |
| extremities, other extremity |
| 170799 Other atherosclerosis of other type of bypass graft(s) of the |
| extremities, unspecified extremity |
| 1739 Peripheral vascular disease, unspecified |

Hyperlipidem ia


| E781 | 2724 | Pure hyperglyceridemia | OTHER AND UNSPECIFIED HYPERLIPIDEMIA |
|---|---|---|---|
| E782 | | Mixed hyperlipidemia | |
| E784 | | Other hyperlipidemia | |
| E785 | | Hyperlipidemia, unspecified | |

Renal dysfunction


| 1 | | | |
|---|---|---|---|
| M1039 | 40413 | Gout due to renal impairment, multiple sites | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| M3214 | 4049 | Glomerular disease in systemic lupus erythematosus | UNSPECIFIED HYPERTENSIVE HEART AND KIDNEY DISEASE |
| M3215 | 40490 | Tubulo-interstitial nephropathy in systemic lupus | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | erythematosus | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | er y thematosus | KIDNEY DISEASE STAGE I THROUGH STAGE IV OR |
| | | | UNSPECIFIED |
| M3504 | 40491 | Sicca syndrome with tubulo-interstitial nephropathy | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| N000 | 40492 | Acute nephritic syndrome with minor glomerular | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | abnormality | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | | KIDNEY DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N001 | 40493 | Acute nephritic syndrome with focal and segmental | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | .0.50 | glomerular lesions | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | giorner didi Tesions | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| 11000 | 4522 | A construction of the difference of the differen | |
| N002 | 4533 | Acute nephritic syndrome with diffuse membranous | EMBOLISM AND THROMBOSIS OF RENAL VEIN |
| | | glomerulonephritis | |
| N003 | 5800 | Acute nephritic syndrome with diffuse mesangial | ACUTE GLOMERULONEPHRITIS WITH LESION OF |
| | | proliferative glomerulonephritis | PROLIFERATIVE GLOMERULONEPHRITIS |
| N004 | 5804 | Acute nephritic syndrome with diffuse endocapillary | ACUTE GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| | | proliferative glomerulonephritis | PROGRESSIVE GLOMERULONEPHRITIS |
| N005 | 5808 | Acute nephritic syndrome with diffuse mesangiocapillary | ACUTE GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
| 11003 | 3000 | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N006 | 5809 | Acute nephritic syndrome with dense deposit disease | ACUTE GLOMERULONEPHRITIS WITH UNSPECIFIED |
| NUUB | 3809 | Acute riepriritic syndrome with dense deposit disease | |
| | | | PATHOLOGICAL LESION IN KIDNEY |
| N007 | 581 | Acute nephritic syndrome with diffuse crescentic | NEPHROTIC SYNDROME |
| | | glomerulonephritis | |
| N008 | 5810 | Acute nephritic syndrome with other morphologic changes | NEPHROTIC SYNDROME WITH LESION OF PROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N009 | 5811 | Acute nephritic syndrome with unspecified morphologic | NEPHROTIC SYNDROME WITH LESION OF MEMBRANOUS |
| | | changes | GLOMERULONEPHRITIS |
| N010 | 5812 | Rapidly progressive nephritic syndrome with minor | NEPHROTIC SYNDROME WITH LESION OF |
| NOTO | 3012 | 1 | |
| | | glomerular abnormality | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N011 | 5813 | Rapidly progressive nephritic syndrome with focal and | NEPHROTIC SYNDROME WITH LESION OF MINIMAL CHANG |
| | | segmental glomerular lesions | GLOMERULONEPHRITIS |
| N012 | 5818 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH OTHER SPECIFIED |
| | | membranous glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N013 | 58181 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME IN DISEASES CLASSIFIED |
| | | mesangial proliferative glomerulonephritis | ELSEWHERE |
| N014 | 58189 | Rapidly progressive nephritic syndrome with diffuse | OTHER NEPHROTIC SYNDROME WITH SPECIFIED |
| 11014 | 20102 | 1 | |
| NO45 | 5040 | endocapillary proliferative glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N015 | 5819 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH UNSPECIFIED PATHOLOGICA |
| | | mesangiocapillary glomerulonephritis | LESION IN KIDNEY |
| N016 | 5820 | Rapidly progressive nephritic syndrome with dense deposit | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | disease | PROLIFERATIVE GLOMERULONEPHRITIS |
| N017 | 5821 | Rapidly progressive nephritic syndrome with diffuse | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | crescentic glomerulonephritis | MEMBRANOUS GLOMERULONEPHRITIS |
| N018 | 5822 | Rapidly progressive nephritic syndrome with other | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| 11010 | 3022 | morphologic changes | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| NO10 | F034 | | |
| N019 | 5824 | Rapidly progressive nephritic syndrome with unspecified | CHRONIC GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| | | morphologic changes | PROGRESSIVE GLOMERULONEPHRITIS |
| N020 | 5828 | Recurrent and persistent hematuria with minor glomerular | CHRONIC GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
| | | abnormality | PATHOLOGICAL LESION IN KIDNEY |
| N021 | 5829 | Recurrent and persistent hematuria with focal and | CHRONIC GLOMERULONEPHRITIS WITH UNSPECIFIED |
| | | segmental glomerular lesions | PATHOLOGICAL LESION IN KIDNEY |
| N022 | 5830 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| INULL | 3030 | · · | |
| | | membranous glomerulonephritis | OR CHRONIC WITH LESION OF PROLIFERATIVE |
| | | Ī | GLOMERULONEPHRITIS |

| N023 | 5831 | Recurrent and persistent hematuria with diffuse mesangial proliferative glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE<br>OR CHRONIC WITH LESION OF MEMBRANOUS<br>GLOMERULONEPHRITIS |
|---|---|---|---|
| N024 | 5832 | Recurrent and persistent hematuria with diffuse endocapillary proliferative glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH LESION OF MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N025 | 5834 | Recurrent and persistent hematuria with diffuse mesangiocapillary glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH LESION OF RAPIDLY PROGRESSIVE GLOMERULONEPHRITIS |
| N026 | 5836 | Recurrent and persistent hematuria with dense deposit disease | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH LESION OF RENAL CORTICAL NECROSIS |
| N027 | 5837 | Recurrent and persistent hematuria with diffuse crescentic glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH LESION OF RENAL MEDULLARY NECROSIS |
| N028 | 5838 | Recurrent and persistent hematuria with other morphologic changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE<br>OR CHRONIC WITH OTHER SPECIFIED PATHOLOGICAL LESION<br>IN KIDNEY |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified morphologic changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE<br>OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN<br>KIDNEY |
| N030 | 5846 | Chronic nephritic syndrome with minor glomerular abnormality | ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS |
| N031 | 5847 | Chronic nephritic syndrome with focal and segmental glomerular lesions | ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLAI (PAPILLARY) NECROSIS |
| N032 | 5848 | Chronic nephritic syndrome with diffuse membranous glomerulonephritis | ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N033 | 5849 | Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis | ACUTE KIDNEY FAILURE UNSPECIFIED |
| N034 | 5851 | Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis | CHRONIC KIDNEY DISEASE STAGE I |
| N035 | 5852 | Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis | CHRONIC KIDNEY DISEASE STAGE II (MILD) |
| N036 | 5853 | Chronic nephritic syndrome with dense deposit disease | CHRONIC KIDNEY DISEASE STAGE III (MODERATE) |
| N037 | 5854 | Chronic nephritic syndrome with diffuse crescentic glomerulonephritis | CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| N038 | 5855 | Chronic nephritic syndrome with other morphologic changes | CHRONIC KIDNEY DISEASE STAGE V |
| N039 | 5856 | Chronic nephritic syndrome with unspecified morphologic changes | END STAGE RENAL DISEASE |
| N040 | 5859 | Nephrotic syndrome with minor glomerular abnormality | CHRONIC KIDNEY DISEASE UNSPECIFIED |
| N041 | 86600 | Nephrotic syndrome with focal and segmental glomerular lesions | UNSPECIFIED INJURY TO KIDNEY WITHOUT OPEN WOUND INTO CAVITY |
| N042 | 86601 | Nephrotic syndrome with diffuse membranous glomerulonephritis | HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE WITHOUT OPEN WOUND INTO CAVITY |
| N043 | 8661 | Nephrotic syndrome with diffuse mesangial proliferative glomerulonephritis | INJURY TO KIDNEY WITH OPEN WOUND INTO CAVITY |
| N044 | | Nephrotic syndrome with diffuse endocapillary proliferative glomerulonephritis | |
| N045 | | Nephrotic syndrome with diffuse mesangiocapillary glomerulonephritis | |
| N046 | | Nephrotic syndrome with dense deposit disease | |
| N047 | | Nephrotic syndrome with diffuse crescentic glomerulonephritis | |
| N048 | | Nephrotic syndrome with other morphologic changes | |
| N049 | | Nephrotic syndrome with unspecified morphologic changes | |
| N050 | | Unspecified nephritic syndrome with minor glomerular abnormality | |
| N051 | | Unspecified nephritic syndrome with focal and segmental glomerular lesions | |
| N052 | | Unspecified nephritic syndrome with diffuse membranous glomerulonephritis | |

| N053 | Unspecified nephritic syndrome with diffuse mesangial |
|---|---|
| | proliferative glomerulonephritis |
| N054 | Unspecified nephritic syndrome with diffuse endocapillary |
| | proliferative glomerulonephritis |
| N055 | Unspecified nephritic syndrome with diffuse |
| | mesangiocapillary glomerulonephritis |
| N056 | Unspecified nephritic syndrome with dense deposit disease |
| N057 | Unspecified nephritic syndrome with diffuse crescentic |
| | glomerulonephritis |
| N058 | Unspecified nephritic syndrome with other morphologic |
| | changes |
| N059 | Unspecified nephritic syndrome with unspecified |
| | morphologic changes |
| N060 | Isolated proteinuria with minor glomerular abnormality |
| N061 | Isolated proteinuria with focal and segmental glomerular |
| 11001 | lesions |
| N062 | Isolated proteinuria with diffuse membranous |
| 11002 | glomerulonephritis |
| N063 | Isolated proteinuria with diffuse mesangial proliferative |
| 11003 | |
| 11054 | glomerulonephritis |
| N064 | Isolated proteinuria with diffuse endocapillary proliferative |
| | glomerulonephritis |
| N065 | Isolated proteinuria with diffuse mesangiocapillary |
| | glomerulonephritis |
| N066 | Isolated proteinuria with dense deposit disease |
| N067 | Isolated proteinuria with diffuse crescentic |
| | glomerulonephritis |
| N068 | Isolated proteinuria with other morphologic lesion |
| N069 | Isolated proteinuria with unspecified morphologic lesion |
| N070 | Hereditary nephropathy, not elsewhere classified with |
| | minor glomerular abnormality |
| N071 | Hereditary nephropathy, not elsewhere classified with focal |
| | and segmental glomerular lesions |
| N072 | Hereditary nephropathy, not elsewhere classified with |
| | diffuse membranous glomerulonephritis |
| N073 | Hereditary nephropathy, not elsewhere classified with |
| 11075 | diffuse mesangial proliferative glomerulonephritis |
| N074 | Hereditary nephropathy, not elsewhere classified with |
| 11074 | |
| NOZE | diffuse endocapillary proliferative glomerulonephritis |
| N075 | Hereditary nephropathy, not elsewhere classified with |
| 11076 | diffuse mesangiocapillary glomerulonephritis |
| N076 | Hereditary nephropathy, not elsewhere classified with |
| | dense deposit disease |
| N077 | Hereditary nephropathy, not elsewhere classified with |
| | diffuse crescentic glomerulonephritis |
| N078 | Hereditary nephropathy, not elsewhere classified with |
| | other morphologic lesions |
| N079 | Hereditary nephropathy, not elsewhere classified with |
| | unspecified morphologic lesions |
| N08 | Glomerular disorders in diseases classified elsewhere |
| N140 | Analgesic nephropathy |
| N141 | Nephropathy induced by other drugs, medicaments and |
| | biological substances |
| N142 | Nephropathy induced by unspecified drug, medicament or |
| | biological substance |
| N143 | Nephropathy induced by heavy metals |
| N144 | Toxic nephropathy, not elsewhere classified |
| N150 | Balkan nephropathy |
| | Other specified renal tubulo-interstitial diseases |
| N158 | Donal tubula interestitial disease |
| N158<br>N159<br>N16 | Renal tubulo-interstitial disease, unspecified Renal tubulo-interstitial disorders in diseases classified |


Chronic liver disease


| K7210 | 5731 | Chronic hepatic failure without coma | HEPATITIS IN VIRAL DISEASES CLASSIFIED ELSEWHERE |
|---|---|---|---|
| K7211 | 5732 | Chronic hepatic failure with coma | HEPATITIS IN OTHER INFECTIOUS DISEASES CLASSIFIED |
| | | | ELSEWHERE |
| K7290 | 5733 | Hepatic failure, unspecified without coma | HEPATITIS UNSPECIFIED |
| K7291 | 5734 | Hepatic failure, unspecified with coma | HEPATIC INFARCTION |
| K730 | 5735 | Chronic persistent hepatitis, not elsewhere classified | HEPATOPULMONARY SYNDROME |
| K731 | 5738 | Chronic lobular hepatitis, not elsewhere classified | OTHER SPECIFIED DISORDERS OF LIVER |
| K732 | 5739 | Chronic active hepatitis, not elsewhere classified | UNSPECIFIED DISORDER OF LIVER |
| K738 | | Other chronic hepatitis, not elsewhere classified | |
| K739 | | Chronic hepatitis, unspecified | |
| K740 | | Hepatic fibrosis | |
| K741 | | Hepatic sclerosis | |
| K742 | | Hepatic fibrosis with hepatic sclerosis | |
| K743 | | Primary biliary cirrhosis | |
| K744 | | Secondary biliary cirrhosis | |
| K745 | | Biliary cirrhosis, unspecified | |
| K7460 | | Unspecified cirrhosis of liver | |
| K7469 | | Other cirrhosis of liver | |
| K750 | | Abscess of liver | |
| K751 | | Phlebitis of portal vein | |
| K752 | | Nonspecific reactive hepatitis | |
| K753 | | Granulomatous hepatitis, not elsewhere classified | |
| K754 | | Autoimmune hepatitis | |
| K7581 | | Nonalcoholic steatohepatitis (NASH) | |
| K7589 | | Other specified inflammatory liver diseases | |
| K759 | | Inflammatory liver disease, unspecified | |
| K760 | | Fatty (change of) liver, not elsewhere classified | |
| K761 | | Chronic passive congestion of liver | |
| K763 | | Infarction of liver | |
| K764 | | Peliosis hepatis | |
| K765 | | Hepatic veno-occlusive disease | |
| K766 | | Portal hypertension | |
| K767 | | Hepatorenal syndrome | |
| K7681 | | Hepatopulmonary syndrome | |
| K7689 | | Other specified diseases of liver | |
| K769 | | Liver disease, unspecified | |
| K77 | | Liver disorders in diseases classified elsewhere | |

<u>Asthma</u>


# Appendix A Comorbid conditions


# Appendix A Nonbiologics

#### **Adalimumab**

This measure categorizes the number of biologic DMARDs into the following categories:

- 0: Up to 1.0 (exclusive). This is the referent category
- 1: From 1.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 3.0 (exclusive).
- >=3: From 3.0 (inclusive) to (any)


Certolizumab pegol

| CERTOLIZUMAB PEGOL |
|--------------------|
| J0718 |

Etanercept


Etanercept

| NDC Brand Name |
|------------------|
| SIMPONI |
| SIMPONI ARIA |
| NDC Generic Name |
| GOLIMUMAB |
| HCPCS |
| J1602 |

# Infliximab


**Abatacept** 

| , marace pr | |
|------------------|-------------------|
| NDC Brand Name | |
| ORENCIA | |
| NDC Generic Name | |
| ABATACEPT | ABATACEPT/MALTOSE |
| HCPCS | |
| C9230 | J0129 |

#### Tocilizumab


#### **Tofacitinib**

This measure categorizes the number of nonbiologic DMARDs into the following categories:

- 0: Up to 1.0 (exclusive). This is the referent category
- 1: From 1.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 3.0 (exclusive).
- >=3: From 3.0 (inclusive) to (any)

| NDC Brand Name |
|---------------------|
| XELJANZ |
| NDC Generic Name |
| TOFACITINIB CITRATE |

#### Auranofin

| 7.00.00.00 | |
|------------------|-------------|
| NDC Brand Name | |
| RIDAURA | |
| NDC Generic Name | |
| AURANOFIN | |
| NDC Drug Code | • |
| 00007487918 | 63032001160 |
| 65483009306 | |

#### Azathioprine

| / Eddinoprinc | |
|------------------|---------------------|
| NDC Brand Name | |
| AZASAN | AZATHIOPRINE SODIUM |
| AZATHIOPRINE | IMURAN |
| NDC Generic Name | |
| AZATHIOPRINE | AZATHIOPRINE SODIUM |

# Cyclophosphamide

| NDC Brand Name | |
|------------------------------|----------------------|
| CYCLOPHOSPHAMIDE | CYTOXAN LYOPHILIZED |
| CYCLOPHOSPHAMIDE MONOHYDRATE | NEOSAR |
| CYTOXAN | NEOSAR FOR INJECTION |
| NDC Generic Name | |
| CYCLOPHOSPHAMIDE | |

#### Cyclosporine

| NDC Brand Name | |
|-----------------------|------------------------|
| CYCLOSPORINE | RESTASIS |
| CYCLOSPORINE MODIFIED | SANDIMMUNE |
| GENGRAF | SANGCYA |
| NEORAL | |
| NDC Generic Name | |
| CYCLOSPORINE | CYCLOSPORINE, MODIFIED |

#### Gold sodium thiomalate

| NDC Brand Name | |
|----------------|-------------|
| AUROLATE | MYOCHRYSINE |

# Appendix A Nonbiologics


# Leflunomide

| NDC Brand Name | |
|------------------|-------------|
| ARAVA | LEFLUNOMIDE |
| NDC Generic Name | |
| LEFLUNOMIDE | |

#### Sulfasalizine

| NDC Brand Name | |
|------------------|------------------|
| AZULFIDINE | SULFASALAZINE DR |
| S.A.S500 | SULFAZINE |
| SULFA DYNE | SULFAZINE EC |
| SULFASALAZINE | |
| NDC Generic Name | |
| SULFASALAZINE | |

# **NSAIDs and Coxibs**

| NDC Generic Name | |
|------------------|------------|
| CELECOXIB | NABUMETONE |
| DIFLUNISAL | NAPROXEN |
| ETODOLAC | OXAPROZIN |
| FLURBIPROFEN | PIROXICAM |
| IBUPROFEN | ROFECOXIB |
| INDOMETHACIN | SULINDAC |
| KETOPROFEN | VALDECOXIB |
| MELOXICAM | |

# Opioids

| NDC Brand Name | |
|--------------------------------|-----------------|
| A-COF DH | LIQUIHISTINE CS |
| ABC COMPOUND W/CODEINE #3 | LORCET |
| ABER-TUSS HC | LORCET 10-650 |
| ABSTRAL | LORCET 10/650 |
| ACAHISTINE | LORCET HD |
| ACETA W/CODEINE | LORCET PLUS |
| ACETAMINOPH-CAFF-DIHYDROCODEIN | LORCIDE |
| ACETAMINOPHEN W-CODEINE | LORTAB |
| ACETAMINOPHEN W/CODEINE | LORTAB ASA |
| ACETAMINOPHEN-CODEINE | LORTUSS EX |
| ACTAGEN-C | LORTUSS HC |
| ACTIFED WITH CODEINE | LYNOX |
| ACTIQ | M-CLEAR |
| ADOL | M-CLEAR JR |
| AIRACOF | M-CLEAR WC |
| ALA-HIST AC | M-END |
| ALAHIST DHC | M-END MAX |
| ALCET | M-END MAX D |
| ALLAY | M-END PE |
| ALLERFRIM W/CODEINE | M-END WC |
| ALLFEN CD | M-GESIC |
| ALLFEN CDX | M-TUSS |
| ALOR | MAGNACET |
| ALPHEN | MAR-COF BP |
| AMACODONE | MAR-COF CG |
| AMAPHEN W/CODEINE NO.3 | MARCOF |

| ANADENIA | MARCECIC |
|---|---|
| AMBENYL | MARGESIC COMPOUND |
| AMBI 5/15/100 | MARGESIC COMPOUND |
| AMBIFED CDV | MARGESIC H |
| AMBIFED_G CD | MARGESIC IMPROVED |
| AMBIFED-G CD AMBIFED-G CDX | MAX HC<br>MAXI-TUSS HC |
| | i |
| AMBOPHEN | MAXI-TUSS HCG |
| AMGENAL<br>AN-ABATE | MAXI-TUSS HCX MAXIDONE |
| ANACIN-3 W/CODEINE | |
| ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE | MAXIFED CD MAXIFED CDX |
| ANAPLEX HD | MAXIFED CDX |
| ANATUSS W/CODEINE | MAXIFED-G CDX |
| ANATOSS W/CODEINE<br>ANEXSIA | MAXIFLU CD |
| ANODYNOS-DHC | MAXIFLU CDX |
| ANOLOR DH-5 | MAXIPHEN CD |
| APOKYN | MAXIPHEN CDX |
| APOMORPHINE HCL | MAXITUSS HC |
| ASA-BUTALB-CAFFEINE-CODEINE | MC COUGH |
| ASCOMP W/CODEINE # 3 | MC JR COUGH |
| ASCOMP WITH CODEINE | MED-HIST |
| ASPIRIN W/CODEINE | MED-HIST-HC |
| ASPIRIN WITH CODEINE | MEDCODIN |
| ASPIRIN WITH CODEINE ASPIRIN-CAFFEINE-DIHYDROCODEIN | MEDICAP HD |
| ASTRAMORPH-PF | MEDICAF IID MEDIPAIN 5 |
| ATROPINE W/DEMEROL | MEDTUSS HD |
| ATUSS EX | MEGAGESIC |
| ATUSS G | MEGAMOR |
| ATUSS HC | MEPERGAN |
| ATUSS HD | MEPERGAN FORTIS |
| ATUSS HS | MEPERIDINE HCL |
| ATUSS HX | MEPERIDINE HCL-0.9% NACL |
| ATUSS MR | MEPERIDINE HCL-NS |
| ATUSS MS | MEPERIDINE HCL/NS |
| ATUSS NX | MEPERIDINE W/PROMETHAZINE |
| AVINZA | MEPERIDINE-PROMETHAZINE |
| AZDONE | MEPERITAB |
| B-TUSS | MEPROZINE |
| BALACET 325 | MESEHIST WC |
| BALTUSSIN | MI-CODE |
| BALTUSSIN HC | MI-DECON |
| BANCAP HC | MINTEX HC |
| BAYCOMINE | MINTUSS EX |
| BAYCOMINE PEDIATRIC | MINTUSS G |
| BAYHISTINE | MINTUSS HC |
| BEXOPHENE | MINTUSS HD |
| BIOTUSSIN AC | MINTUSS MR |
| BIOTUSSIN DAC | MINTUSS MS |
| BIPHETANE-DC | MINTUSS NX |
| BITEX | MONTE-G HC |
| BPM PE HC | MONTEFLU HC |
| BROM-CORT-DC | MORPHINE SULF/D5W |
| BROMANATE DC | MORPHINE SULF/NS |
| BROMANATE-DC | MORPHINE SULFATE |
| BROMANYL | MORPHINE SULFATE CONCENTRATE |
| BROMAREST DC | MORPHINE SULFATE CR |
| BROMATANE-DC | MORPHINE SULFATE ER |
| BROMCOMP HC | MORPHINE SULFATE IN DEXTROSE |
| BROMODIPHENHYDRAMINE HCL | MORPHINE SULFATE INJECTION |
| BROMODIPHENHYDRAMINE W/CODEINE | MORPHINE SULFATE SELECT-A-JET |
| | _ |
| BROMOTUSS W/CODEINE | MORPHINE SULFATE-0.9% NACL |

| BROWENIEW HD | MODDIUME CITIENTE (DEM |
|--------------------------------|------------------------|
| BROMPHENEX HD | MORPHINE SULFATE/NS |
| BROMPHENIRAMINE DC | MORPHINE SULFATE/NS |
| BROMPHENIRAMINE-DC | MS CONTIN |
| BROMPHENIRAMINE-DC W/CODEINE | MS/L |
| BROMPHENIRAMINE-HYDROCOD-PSE | MS/S |
| BROMPLEX HD | MSIR |
| BRON-TUSS | MULTI-HIST CS |
| BRONKISAN A/C | MYBANIL |
| BRONTEX | MYCI-GC |
| BROVEX CB | MYGRANOL W/CODEINE #3 |
| BROVEX CBX | MYHYDROMINE |
| BROVEX HC | MYHYDROMINE PEDIATRIC |
| BROVEX PB C | MYPHETANE DC |
| BROVEX PB CX | MYTUSSIN AC |
| BUTALB-ACETAMINOPH-CAFF-CODEIN | MYTUSSIN DAC |
| BUTALB-CAFF-ACETAMINOPH-CODEIN | NALDECON-CX ADULT |
| BUTALBITAL COMPOUND W/CODEINE | NALEX |
| BUTALBITAL COMPOUND-CODEINE | NALEX AC |
| BUTALBITAL-CAFF-APAP-CODEINE | NALEX DH |
| BUTALBITAL/CAFF/APAP/CODEINE | NARCOF |
| BUTINAL W/CODEINE #3 | NARIZ HC |
| C-TUSSIN | NARVOX |
| CALCIDRINE | NASATUSS |
| CALCIUM IODIDE W/CODEINE | NASOTUSS |
| , | |
| CANGES-HC | NAZARIN HC |
| CANGES-HC NR | NEO AC |
| CANGES-XP | NEO HC |
| CAPCOF | NORCET |
| CAPITAL W-CODEINE | NORCET 7.5MG |
| CAPITAL W/CODEINE | NORCO |
| CARISOPRODOL COMPOUND-CODEINE | NOTUSS |
| CARISOPRODOL-ASPIRIN-CODEINE | NOTUSS AC |
| CENTUSSIN DHC | NOTUSS DC |
| CETA-PLUS | NOTUSS PD |
| CGU WC | NOTUSS-FORTE |
| CHEMDAL | NOTUSS-NX |
| CHEMERGAN W/CODEINE | NOTUSS-NXD |
| CHERACOL | NOTUSS-PE |
| CHERATUSSIN AC | NOVADYNE |
| CHERATUSSIN DAC | NOVADYNE DH |
| CHLORPHEN HD | NOVAGEST |
| CHLORPHENIRAMINE-CODEINE | NOVAGEST DH |
| CLEARTUSS DH | NOVAHISTINE |
| CO-GESIC | NOVAHISTINE DH |
| CO-HISTINE | NOVASUS |
| CO-HISTINE DH | NUCOCHEM |
| COASTALDYNE | NUCODINE SYR |
| COCET | NUCOFED |
| COCET PLUS | NUCOTUSS |
| CODACA NO.3 | NUDAL-HD |
| CODACED | NUMORPHAN |
| CODAL DI | OMS |
| CODAMINE | ONCET |
| CODAMINE | ONCET 5 |
| CODAMINE PEDIATRIC | ONCET 7 |
| CODAPHEN | ONSOLIS |
| CODAR AR | OPANA |
| CODAR D | OPANA ER |
| CODAR GF | ORAMORPH SR |
| CODEFEN | ORGADIN-TUSS |
| CODEGEST | OXECTA |
| CODEINE COUGH SYRUP | OXYCODONE CONCENTRATE |
| CODEINE COOGH SINOI | |

| CODEINE PHOSPHATE | OXYCODONE HCL |
|--------------------------------|---------------------------------------------|
| CODEINE SULFATE | OXYCODONE HCL ER |
| CODEINE-GUAIFENESIN | OXYCODONE HCL-ACETAMINOPHEN |
| CODEINE/PHENYLPROP/GUAIFENESIN | OXYCODONE HCL-ASPIRIN |
| CODEMINE | OXYCODONE HCL-IBUPROFEN |
| CODICLEAR DH | OXYCODONE HYDROCHLORIDE |
| CODIMAL DH | OXYCODONE W/ACETAMINOPHEN |
| CODIMAL PH | OXYCODONE W/ASPIRIN |
| CODITUSS DH | OXYCODONE W/ASPIRIN HALF-STR |
| CODOTUSS | OXYCODONE-ACETAMINOPHEN |
| COLDCOUGH | OXYCODONE-ASPIRIN |
| COLDCOUGH EXP | OXYCODONE/APAP |
| COLDCOUGH HC | OXYCONTIN |
| COLDCOUGH HCM | OXYFAST |
| COLDCOUGH PD | OXYIR |
| COLDCOUGH XP | OXYMORPHONE HCL |
| COLDTUSS | OXYMORPHONE HCL ER |
| COLREX COMPOUND | P-EPD HCL/HCOD BT/CARBINOX |
| COMBUNOX | P-EPHED HCL/HYDROCOD BIT/CP |
| COMTUSSIN HC | P-TUSS |
| CONDASIN | P-TUSS D |
| CONEX W/CODEINE | P-V-TUSSIN |
| CONZIP | PALLADONE |
| COPAN | PANACET |
| COPHENE XP | PANADOL W/CODEINE NO.3 |
| COPHENE-S | PANADOL W/CODEINE NO.4 |
| CORDRON-HC | PANASAL |
| COTAB A | PANCET |
| COTAB AX | PANCOF |
| COTABFLU | PANCOF EXP |
| COTUSS EX | PANCOF HC |
| COTUSS HD | PANCOF PD |
| COTUSS MS | PANCOF XP |
| COTUSS-V | PANLOR |
| COUGHTUSS | PANLOR DC |
| CPB WC | PANLOR SS |
| CRANTEX HC | PAPA-DEINE NO.4 |
| CYCOFED | PC-CAP |
| CYNDAL | PEDIACOF |
| CYTUSS HC | PEDIATEX HC |
| CYTUSS-HC | PEDITUSS |
| D-TANN HC | PERCOCET |
| DAMASON-P | PERCODAN |
| DARVOCET ALGO | PERCODAN DEMI |
| DARVOCET N 50 | PERCOLONE |
| DARVOCET-N 50 | PERLOXX |
| DARVON | PHANATUSS HC |
| DARVON COMPOUND 33 | PHEN/CHLOR HC |
| DARVON COMPOUND GE | PHENA-HC |
| DARVON N | PHENAPHEN W/CODEINE |
| DARVON-N | PHENDACOF PLUS |
| DAZIDOX | |
| DE-CHLOR G | PHENERGAN VC W/CODEINE |
| DE-CHLOR HC | PHENERGAN W/CODEINE |
| DE-CHLOR HD | PHENERGAN W/CODEINE PHENERGAN WITH CODEINE |
| DE-CHLOR MR | |
| DE-CHLOR NX DECOHISTINE | PHENFLU CD PHENFLU CDX |
| DECOHISTINE DH DECONAMINE CX | PHENHIST PHENYLCODONE PEDIATRIC |
| DECONGEST | PHENYLEODONE PEDIATRIC PHENYLEPH-HCOD BT-CP |
| DECTUSS C | PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD |
| טנכוטטכ | FIILN ILLE NAME NO |

| DELHISTINE CS | PHENYLHISTINE |
|--------------------------|--------------------------------|
| DEMEROL | PHENYLHISTINE DH |
| DEPODUR | PHENYLPROP/COD/BR-PHENIRAMINE |
| DESPEC-EXP | PHENYLPROPANOLAMINE DC |
| DESPEC-PD | PHENYLPROPANOLAMINE/HYDROCODON |
| DESPEC-PDC | PHRENILIN W/CAFFEINE & CODEINE |
| DETUSS | PHRENILIN-CAFFEINE-CODEINE |
| DETUSSIN | PLURATUSS |
| DEX-TUSS | PNAP |
| DEXPHEN W-C | PNEUMOTUSSIN |
| DIABETIC TUSSIN C | PNEUMOTUSSIN HC |
| DIHIST DH | POLY CS |
| DIHISTINE DILICTINE DIL | POLY HIST DHC POLY HIST HC |
| DIHISTINE DH | POLY HIST NC |
| DIHYDRO-CP | |
| DIHYDRO-GP | POLY-USTINE |
| DIHYDRO-PE | POLY-HISTINE CC |
| DIHYDROCODEINE COMP MOD | POLY-HISTINE CS |
| DIHYDROCODEINE COMPOUND | POLY TUSSIN |
| DIHYDROCODEINE-BPM-PE | POLY-TUSSIN AC |
| DIHYDROXCODEINE COMPOUND | POLY-TUSSIN D |
| DILAUDID | POLY-TUSSIN DHC |
| DILAUDID STRIP PACKS | POLY-TUSSIN EX |
| DILAUDID-5 | POLY-TUSSIN HD |
| DILAUDID-HP | POLY-TUSSIN XP |
| DIMETANE-DC | POLYGESIC |
| DOLACET | POLYTINE CS |
| DOLAGESIC | POT GUAIACO-HYDROCODONE BIT |
| DOLENE | PP-CAP |
| DOLENE AP-65 | PRIMALEV |
| DOLENE COMPOUND-65 | PRIMLEV |
| DOLFEN | PRO POX 65 |
| DOLO PAP | PRO-CLEAR |
| DOLO-PAP | PRO-CLEAR AC |
| DOLOREX FORTE | PRO-CLEAR CAPS |
| DOLPHEN | PRO-COF |
| DONATUSS DC | PRO-COF D |
| DONATUSSIN DC | PRO-RED |
| DONATUSSIN MAX | PRO-RED AC |
| DORAPHEN-65 | PROCET |
| DOXAPAP N-100 | PROLEX DH |
| DRITUSS HD | PROMETHAZINE VC W/CODEINE |
| DROCON-CS | PROMETHAZINE VC-CODEINE |
| DROTUSS | PROMETHAZINE W/CODEINE |
| DROTUSS-CP | PROMETHAZINE-CODEINE |
| DUOCET | PROPACET |
| DUOHIST DH | PROPACHEM |
| DURADAL | PROPACHEM PEDIATRIC |
| DURADAL HD | PROPAIN HC |
| DURADAL HD PLUS | PROPOXACET-N 100 |
| DURADYNE DHC | PROPOXYPHENE HCL |
| DURAGANIDIN NR | PROPOXYPHENE HCL COMPOUND |
| DURAGESIC | PROPOXYPHENE HCL W/APAP |
| DURAMORPH | PROPOXYPHENE HCL-ACETAMINOPHEN |
| DURATUSS HD | PROPOXYPHENE NAP-ACETAMINOPHEN |
| DYNATUSS DF | PROPOXYPHENE NAPSYLATE |
| DYNATUSS HC | PROPOXYPHENE NAPSYLATE W/APAP |
| DYNATUSS HCG | PROPOXYPHENE NAPSYLATE-APAP |
| DYNEX HD | PROTEX |
| DYTAN-HC | PROTEX D |
| E-LOR | PROTUSS |
| ED TUSS HC | PROTUSS-D |
| - | |

| ED-TLC | PROVAL NO.3 |
|----------------------------|-------------------------------|
| EFASIN | PSE BPM HD |
| EFASIN-HD | PSEUDATEX HC |
| EMBEDA | PSEUDOEPHEDRINE W/CODEINE |
| EMCODEINE NO.3 | PSEUDOEPHEDRINE W/HYDROCODONE |
| EMCODEINE NO.4 | PSEUDOEPHEDRINE-CODEINE |
| EMPIRIN W/CODEINE | Q-V TUSSIN |
| EMPRACET W/CODEINE NO.3 | QUAL-TUSSIN DC |
| EMPRACET W/CODEINE NO.4 | QUALA-HC |
| ENDACOF | QUINDAL |
| ENDACOF AC | QUINDAL-HD |
| ENDACOF-C | QUINTEX HC |
| ENDACOF-C ENDACOF-DC | RELACON-HC |
| ENDACOF-DH | RELACON-HC NR |
| ENDACOF-HC | RELACIN-HC NK |
| ENDACOF-PLUS | RELASIN-HCX |
| ENDACOF-XP | RELATUSS HC |
| ENDAGEN-HD | RELCOF C |
| ENDAL | REPREXAIN |
| ENDAL CD | RESCUDOSE |
| ENDAL HD | REX-A-HIST |
| ENDAL-HD | REZIRA |
| ENDAL-HD PLUS | RHINACON DH |
| ENDOCET | RID-A-PAIN W/CODEINE |
| ENDOCODONE | RINDAL HD |
| ENDODAN | RINDAL HD PLUS |
| ENDOTUSS | RINDAL HPD |
| ENPLUS-HD | RMS-SUPPOSITORY |
| ENTEX HC | RO-CET-N 100 |
| ENTUSS | ROBAFEN AC |
| ENTUSS-D | ROBAFEN-DAC |
| ESGIC W/CODEINE | ROBICHEM AC |
| ETH-OXYDOSE | ROBITUSSIN A-C |
| EXALGO | ROBITUSSIN-DAC |
| EXCOF | ROGESIC #3 |
| EXCOF-SF | ROMILAR AC |
| EXECLEAR | ROXANOL |
| EXECLEAR-C | ROXANOL SR |
| EXECOF-XP | ROXANOL UD |
| EXETUSS-HC | ROXANOL-T |
| EXTENDRYL HC | ROXICET |
| FARBITAL W/CODEINE #3 | ROXICODONE |
| FEBRIDYNE | ROXICODONE INTENSOL |
| FENTANYL | ROXIPRIN |
| FENTANYL BASE | RYBIX ODT |
| FENTANYL CITRATE | RYDEX |
| FENTANYL CITRATE-0.9% NACL | RYNA-C |
| FENTANYL CITRATE-D5W | RYNA-CX |
| FENTANYL CITRATE-NS | RYZOLT |
| FENTANYL CITRATE-NS | S-T FORTE 2 |
| FENTANYL ORALET | SENEFEN III |
| FENTANYL W/DROPERIDOL | SIMUC-HD |
| FENTANYL WITH DROPERIDOL | SINODEINE |
| FENTANYL-BUPIVACAINE-NS | SK-65 |
| FENTANYL-ROPIVACAINE-NS | SK-65 APAP |
| FENTANYL/NS | SK-65 COMPOUND |
| FENTORA | SK-APAP W/CODEINE |
| FENTUSS | SK-OXYCODONE W/ACETAMINOPHEN |
| FIORICET W/CODEINE | SK-OXYCODONE W/ASPIRIN |
| FIORICET WITH CODEINE | SOMA COMPOUND W/CODEINE |
| FIORINAL W/CODEINE #3 | SOMA COMPOUND WITH CODEINE |
| FIORINAL WITH CODEINE #3 | SPEN-HISTINE |

| | I |
|---|---|
| FIORMOR W/CODEINE #3 | STAGESIC |
| FIORTAL W/CODEINE #3 | STAGESIC-10 |
| FLUTUSS HC | STATUSS |
| FLUTUSS XP | STATUSS GREEN |
| G-TUSS | STERAPHEN W/CODEINE |
| GANI-TUSS NR | STOPAYNE |
| GECIL | SU-TUSS HD |
| GENAGESIC<br>GENECOF-HC | SUBLIMAZE<br>SUBSYS |
| | SUDATUSS-2 |
| GENECOF-XP<br>GENTEX HC | SUDATUSS-SF |
| GESIC-5 | SUTTAR-2 |
| GESIC-5<br>GESIC-HD | |
| GESTUSS-HC | SUTTAR-SF<br>SYMTAN |
| GILTUSS HC | SYMTAN A |
| GILTUSS PED-C | SYNALGOS-DC |
| GLYDEINE | SYNGESIC DC |
| GUA C | SYNGESIC-DC |
| GUAPC | T-GESIC |
| GUAIATUSSIN AC | T-GESIC FORTE |
| GUAIFEN-C | THERACODOPHEN-325 |
| GUAIFENESIN A.C. | THERACODOPHEN-650 |
| GUAIFENESIN A.C. | THERACODOPHEN-LOW-90 |
| GUAIFENESIN DAC | THERATRAMADOL-60 |
| GUAIFENESIN NR | THERATRAMADOL-90 |
| GUAIFENESIN W-CODEINE | TL-HIST CD |
| GUAIFENESIN W-CODEINE | TL-HIST CM |
| GUAIFENESIN-CODEINE | TOURO HC |
| GUAIFENESIN-P-EPHEDRINE-COD | TRAMADOL HCL |
| GUAIFENESIN-PHENYLEPHRINE-HCOD | TRAMADOL HCL ER |
| GUAIFENESIN/CODEINE PHOSPHATE | TRAMADOL HCL-ACETAMINOPHEN |
| · | |
| GUAIFENESIN/P-EPHED HCL/HCOD | TREZIX |
| GUAIFENESIN/P-EPHED HCL/HCOD<br>GUAIFENESIN/P-EPHEDRINE/COD | TREZIX TRI-VENT HC |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC | TREZIX TRI-VENT HC TRIACIN C |
| GUAIFENESIN/P-EPHED HCL/HCOD<br>GUAIFENESIN/P-EPHEDRINE/COD | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE TRICOF |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS IN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE-D | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF PD |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN AC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF PD TRIDAL |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF PD TRIDAL TRIDAL TRIDAL |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-DAC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODE W/CODEINE TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODE W/CODEINE TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIHIST-CS |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-DAC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI | TREZIX TRI-VENT HC TRIACIN C TRIAGIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODE W/CODEINE TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-DAC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM | TREZIX TRI-VENT HC TRIACIN C TRIAGIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF EXP TRICOF PD TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPOSED W/CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC | TREZIX TRI-VENT HC TRIACIN C TRIAGIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-DAC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS | TREZIX TRI-VENT HC TRIACIN C TRIAGIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPOLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS | TREZIX TRI-VENT HC TRIACIN C TRIAGEN WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICOPE TRICOF TRICOF EXP TRICOF EXP TRICOF TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPOLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICOPE TRICOF TRICOF TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRYCET TRYMINE CG |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HISTI-PLUS HISTAFED-C HISTEX HC HISTINEX HC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICOPE TRICOF TRICOF TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HISTI-PLUS HISTAFED-C HISTINEX HC HISTINEX PV | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIPOSED W/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS AC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN-AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HISTI-PLUS HISTAFED-C HISTEX HC HISTINEX PV HISTUSS HC | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPOLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD GUAITUSSIN AC GUAITUSSIN DAC GUAITUSSIN DAC GUAL-CO GUAPETEX HC GUIADEX DH GUIAOLEX HC GUIATUSS AC GUIATUSS DAC GUIATUSS DAC GUIATUSSIN DAC GUIATUSSIN W/CODEINE H-C TUSSIVE H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTINEX HC HISTINEX PV HISTUSSIN D | TREZIX TRI-VENT HC TRIACIN C TRIACIN-C TRIAFED WITH CODEINE TRIAMINIC DH TRIAMINIC W/CODEINE TRIANT-HC TRICODE AR TRICODE GF TRICODENE W/CODEINE TRICOF EXP TRICOF EXP TRICOF EXP TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFED-C TRIPOSED W/CODEINE |

| LIDD FAID | TUCC DC |
|---|---|
| HPR END | TUSS-DS |
| HY-5 | TUSS-ES |
| HY-KXP | TUSS-HC |
| HY-PHEN | TUSS-PD |
| HYCET | TUSS-S |
| HYCO-PAP | TUSSADUR-HD |
| HYCODAN | TUSSAFED-HC |
| HYCODAPHEN | TUSSAFED-HCG |
| HYCOFED | TUSSAR-2 |
| HYCOGESIC | TUSSCOUGH DHC |
| HYCOMAL DH | TUSSCOUGH HC |
| HYCOMED | TUSSEND |
| HYCOMINE | TUSSHISTINE CS |
| HYCOMINE COMPOUND | TUSSI-ORGANIDIN NR |
| HYCOPHEN | TUSSI-ORGANIDIN-S NR |
| HYCOSIN | TUSSICAPS |
| HYCOTAB | TUSSICLEAR DH |
| HYCOTUSS | TUSSIDEN C |
| HYDEX PD | TUSSIDIN NR |
| HYDONE | TUSSIGON |
| HYDRO GP | TUSSIN AC |
| HYDRO PC II | TUSSINAL 12 |
| HYDRO PRO | TUSSINATE |
| HYDRO PRO D | TUSSIONEX |
| HYDRO-DP | TUSSIREX |
| HYDRO-PC | TUSSIVE HC |
| HYDRO-PC II PLUS | TUSSO-C |
| HYDRO-PROPANOLAMINE PEDIATRIC | TUSSO-DF |
| HYDRO-TUSS | TUSSO-HC |
| HYDRO-TUSSIN DHC | TUSSPLEX |
| HYDRO-TUSSIN EXP | TY-PAP W/CODEINE |
| LIVE DO TUCCINI IIC | TV TAB IN ICODENIE |
| HYDRO-TUSSIN HC | TY-TAB W/CODEINE |
| HYDRO-TUSSIN HD | TYLAGESIC 3 |
| HYDRO-TUSSIN HD<br>HYDRO-TUSSIN HG | TYLAGESIC 3 TYLENOL W/CODEINE |
| HYDRO-TUSSIN HD<br>HYDRO-TUSSIN HG<br>HYDRO-TUSSIN XP | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCOT HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BITARTRATE | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCOT HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCOT HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE BT-HOMATROPINE MBR | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAME ULTRAM ER |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND HYDROCODONE COMPOUND HYDROCODONE CF | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRAGESIC ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE GF | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC |
| HYDRO-TUSSIN HD HYDRO-TUSSIN HG HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE FA | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF |
| HYDRO-TUSSIN HD HYDRO-TUSSIN YP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP |
| HYDRO-TUSSIN HD HYDRO-TUSSIN YP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE GF HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE HD HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN | TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV |
| HYDRO-TUSSIN HD HYDRO-TUSSIN YP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BITARTRATE HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN | TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.4 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-TRICOF HC |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GF HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE FA HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP | TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL CODEINE NO.4 TYLENOL-CODEINE NO.4 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-TRICOF HC VANACET |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GF HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GF HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-TRICOF HC VANACOF CD |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GOMPOUND HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-TRICOF HC VANACET VANACOR |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCODONE HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GOMPOUND HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOR VANEX GRAPE VANEX HD |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GOMPOUND HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/FHENYLPROP HYDROCODONE GF HYDROCODONE W/FHENYLPROP HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE MBR | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCOT HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GOMPOUND HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/FHENYLPROP HYDROCODONE W/FHENYLPROP HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-BUPROFEN HYDROCODONE-BUPROFEN HYDROCODONE-POT GUAIACOSULFON | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCET HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-BUPROFEN HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BT-HOMATROPINE MBR HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/PHENYLPROP HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-BUPROFEN HYDROCODONE-BUPROFEN HYDROCODONE-BUPROFEN HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/ACETAMINOPHEN | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF UNI-COF UNI-COF UNI-LEV UNI-TRICOF HC VANACOR VANACOR VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET |
| HYDRO-TUSSIN HD HYDRO-TUSSIN XP HYDROCOT HYDROCOD BIT-PHENYLEPHRINE-CP HYDROCOD-CPM-PSEUDOEPHEDRINE HYDROCOD/CARBINOX/PSEUDOEPHED HYDROCODONE HYDROCODONE BIT-HOMATROPINE MB HYDROCODONE BIT-IBUPROFEN HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE BIT-HOMATROPINE MBR HYDROCODONE GOMPOUND HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/FHENYLPROP HYDROCODONE W/FHENYLPROP HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-BUPROFEN HYDROCODONE-BUPROFEN HYDROCODONE-POT GUAIACOSULFON | TYLAGESIC 3 TYLENOL W/CODEINE TYLENOL W/CODEINE NO.2 TYLENOL W/CODEINE NO.3 TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 TYLENOL-CODEINE NO.4 TYLOX UGESIC ULTRACET ULTRAGESIC ULTRAM ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE |

| LIVER OCCUPANTE / DUTANI / DRODANIO LANGUA | Lucopiu |
|---|---|
| HYDROCODONE/PHENYLPROPANOLAMIN | VICODIN |
| HYDROCOF-HC | VICODIN ES |
| HYDROFED | VICODIN HP |
| HYDROGESIC | VICODIN TUSS |
| HYDROMET | VICOPROFEN |
| HYDROMINE LIVER DAMES DE DIATRIC | VIHISTINE |
| HYDROMINE PEDIATRIC | VIRTUSSIN AC |
| HYDROMORPHONE ER | VISVEX HC |
| HYDROMORPHONE HCL | VITAPAP W/CODEINE |
| HYDROMORPHONE HCL INJECTION | VITUSSIN |
| HYDROMORPHONE HCL-D5W | VITUZ |
| HYDROMORPHONE HCL-NS | VOPAC |
| HYDROMORPHONE HCL/NS | W/W-HISTINE |
| HYDROMORPHONE HYDROCHLORIDE | WELL-TUSS HD |
| HYDROMORPHONE-BUPIVACAINE | WELLTUSS EXP |
| HYDROMORPHONE-BUPIVACAINE-NS | WELLTUSS HC |
| HYDROMORPHONE/BUPIVACAINE | WYGESIC |
| HYDRON CP | XARTEMIS XR |
| HYDRON EX | XODOL 10-300 |
| HYDRON KGS | XODOL 10/300 |
| HYDRON PSC | XODOL 5-300 |
| HYDROPANE | XODOL 7.5-300 |
| HYDROPHEN | XOLOX |
| HYDROPHEN PEDIATRIC | XPECT-HC |
| HYDROPHENE DH | XYLON 10 |
| HYDROSTAT | Z-COF HC |
| HYPHED | Z-COF HCX |
| HYPHEN-HD | Z-TUSS 2 |
| HYTAN | Z-TUSS AC |
| IBUDONE | Z-TUSS E |
| IDENAL W/CODEINE | ZAMICET |
| INFUMORPH | ZERLOR |
| INNOVAR | ZHIST |
| INNOVAR<br>IODAL HD | ZHIST ZODRYL AC 25 |
| INNOVAR IODAL HD IOFEN-C NF | ZHIST ZODRYL AC 25 ZODRYL AC 30 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLLYL W/CODEINE J-CET | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLLYL W/CODEINE | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 40 ZODRYL DAC 40 ZODRYL DAC 50 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 40 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 60 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-TAN D HC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 35 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 40 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 60 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-TAN D HC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 35 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 30 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 30 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF JAYCOF-HC JAYCOF-XP KADIAN KG-DAL HD | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 30 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 35 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-XP KADIAN | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 50 ZODRYL DEC 50 ZODRYL DEC 60 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF JAYCOF-HC JAYCOF-XP KADIAN KG-DAL HD | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 50 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-XP KADIAN KG-DAL HD KG-DAL HD PLUS | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 60 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 50 ZODRYL DEC 50 ZODRYL DEC 60 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-HC JAYCOF-XP KADIAN KG-DAL HD KG-DAL HD PLUS KG-FED | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 25 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 40 ZODRYL DEC 60 ZODRYL DEC 60 ZODRYL DEC 60 ZODRYL DEC 80 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-KP KADIAN KG-DAL HD KG-DAL HD PLUS KG-FED KG-FED PEDIATRIC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 80 ZODRYL DEC 80 ZODRYL DEC 80 ZODRYL DEC 80 ZODRYL DEC 80 |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-KP KADIAN KG-DAL HD KG-DAL HD KG-FED PEDIATRIC KG-TUSS HD | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 60 ZODRYL DEC 80 ZODRYL DEC 80 ZOHYDRO ER ZOLVIT |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-HC JAYCOF-XP KADIAN KG-DAL HD PLUS KG-FED KG-FED PEDIATRIC KG-TUSSIN | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 36 ZODRYL DEC 36 ZODRYL DEC 35 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 80 ZODRYL DEC 80 ZOHYDRO ER ZOLVIT ZOTEX-C |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-NP KADIAN KG-DAL HD KG-DAL HD PLUS KG-FED KG-FED PEDIATRIC KG-TUSSIN KGS-HC | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 36 ZODRYL DEC 36 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 50 ZODRYL DEC 80 ZODRYL DEC 80 ZOHYDRO ER ZOLVIT ZOTEX-C ZOTEX-HC |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-HC JAYCOF-HC JAYCOF-XP KADIAN KG-DAL HD PLUS KG-FED PEDIATRIC KG-TUSSIN KGS-HC KWELCOF | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DAC 80 ZODRYL DEC 25 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 30 ZODRYL DEC 40 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 80 ZODRYL DEC 80 ZOHYDRO ER ZOLVIT ZOTEX-C ZOTEX-HC |
| INNOVAR IODAL HD IOFEN-C NF IOPHEN IOPHEN C-NR IOPHEN-C NR IOTUSSIN D IOTUSSIN HC ISOBUTAL W/CODEINE ISOLIN W/CODEINE ISOLLYL W/CODEINE J-CET J-COF DHC J-MAX DHC J-TAN D HC JAYCOF-JAYCOF-HC JAYCOF-HC JAYCOF-AP KADIAN KG-DAL HD PLUS KG-FED PEDIATRIC KG-TUSSIN KG-HC KWELCOF LAZANDA | ZHIST ZODRYL AC 25 ZODRYL AC 30 ZODRYL AC 35 ZODRYL AC 40 ZODRYL AC 50 ZODRYL AC 60 ZODRYL AC 80 ZODRYL DAC 25 ZODRYL DAC 35 ZODRYL DAC 35 ZODRYL DAC 30 ZODRYL DAC 40 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 50 ZODRYL DAC 60 ZODRYL DAC 80 ZODRYL DEC 25 ZODRYL DEC 35 ZODRYL DEC 35 ZODRYL DEC 30 ZODRYL DEC 40 ZODRYL DEC 40 ZODRYL DEC 50 ZODRYL DEC 80 ZODRYL DEC 80 ZOHYDRO ER ZOLVIT ZOTEX-C ZOTEX-HC ZTUSS ZTUSS ZT |

| [. <del>-</del> | |
|---|---|
| LEXUSS 210 | ZYMINE HC |
| LIQUICET | ZYRPHEN-HC |
| LIQUICOUGH HC | |
| NDC Generic Name | MEDEDIDINE LICE IN O.O. (CODILINA CITI ODIDE |
| BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE | MEPERIDINE HCL IN 0.9 % SODIUM CHLORIDE |
| BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE | MEPERIDINE HCL/PF |
| BROMPHENIRAMINE MALEATE/PHENYLEPHRINE | MEPERIDINE HCL/PROMETHAZINE HCL |
| · | MORPHINE SULFATE IN O.0 % SODIUM CHI ORIDE |
| BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE | MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE |
| CHLORCYCLIZINE HCL/CODEINE PHOSPHATE | MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF |
| CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE | MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER |
| CHLORCYCLIZINE HCL/PRENTLEPHRINE HCL/CODEINE PHOSPHATE | MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF |
| CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE | MORPHINE SULFATE/DEXTROSE 5% WATER/FF MORPHINE SULFATE/NALTREXONE HCL |
| CHLORPHENIRAMINE MALEATE/CODEINE | MORPHINE SULFATE/PF |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE | OXYCODONE HCL |
| CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE | OXYCODONE HCL/ACETAMINOPHEN |
| CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN | OXYCODONE/ASPIRIN |
| CODEINE PHOSPHATE/PYRILAMINE MALEATE | OXYMORPHONE HCL |
| CODEINE SULFATE | PHENYLEPHRINE HCL/CODEINE PHOSPHATE |
| CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLEPHRINE HCL/CODEINE |
| CODEINE/CALCIUM IODIDE | PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN |
| DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE | PHENYLEPHRINE |
| DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE | PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE |
| DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE | PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE/POTASSIUM |
| DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE | PHENYLEPHRINE HCL/CODEINE/PYRILAMINE |
| DIHYDROCODEINE BITARTRATE/GUAIFENESIN | PHENYLEPHRINE HCL/DIHYDROCODEINE BITARTRATE |
| DIHYDROCODEINE/ASPIRIN/CAFFEINE | PHENYLEPHRINE HCL/DIHYDROCODEINE |
| DIPHENHYDRAMINE HCL/PHENYLEPHRINE HCL/CODEINE | PHENYLEPHRINE HCL/DIHYDROCODEINE |
| FENTANYL | PHENYLEPHRINE HCL/PPA |
| FENTANYL FENTANYL CITRATE | PHENYLEPHRINE HCL/PPA PHENYLEPHRINE TANNATE/HYDROCODONE |
| FENTANYL CITRATE | PHENYLEPHRINE TANNATE/HYDROCODONE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE HCL/ASPIRIN/CAFFEINE PROPOXYPHENE NAPSYLATE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE HCL/ASPIRIN/CAFFEINE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOSYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ASPIRIN | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ASPIRIN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ASPIRIN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ASPIRIN/CAFFEINE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DIHYDROCODONE BITARTRATE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ASPIRIN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DIHYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE/IBUPROFEN | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DIHYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/HOMATROPINE METHYLBROMIDE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE/IBUPROFEN HYDROMORPHONE HCL | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DIHYDROCODONE BITARTRATE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/HOMATROPINE METHYLBROMIDE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE/IBUPROFEN HYDROMORPHONE HCL HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DIHYDROCODONE BITARTRATE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE HCL IN 0.9 % SODIUM CHLORIDE HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DIHYDROCODONE BITARTRATE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE TANNATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/DHYDROCODEINE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HUDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE TANNATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE HUDROFEN HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL/BUPIVACAINE HCL IN 0.9% SODIUM | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PSEUDOEPHEDRINE/PSEUDOEPHEDRINE HCL/CODEINE BT PYRILAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/PF FENTANYL CITRATE/BODIUM CHLORIDE PF HYDROCODONE BITATTATE/CHLORPHENIRAMINE TANNATE HYDROCODONE HOLL IN 0.9 % SODIUM CHLORIDE PF HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL/PF | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE HCL/CODEINE PROPOXYPHENE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PSEUDOEPHEDRINE/PSEUDOEPHEDRINE HCL/CODEINE BT PYRILAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE TRAMADOL HCL |
| FENTANYL CITRATE FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM FENTANYL CITRATE/DEXTROSE 5% WATER/PF FENTANYL CITRATE/DROPERIDOL FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/PF FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/HYDROCODONE BITARTRATE GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE GUAIFENESIN/PHENYLPROPANOLAMINE GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE GUAIFENESIN/PSEUDOEPHEDRINE HYDROCODONE BITARTRATE HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/ACETAMINOPHEN HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE HYDROCODONE BITARTRATE/CHLORPHENIRAMINE TANNATE HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE HYDROCODONE HOLL HYDROMORPHONE HCL HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF HYDROMORPHONE HCL/BUPIVACAINE HCL IN 0.9% SODIUM | PHENYLEPHRINE TANNATE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE PROMETHAZINE HCL/CODEINE PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL/ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE PSEUDOEPHEDRINE HCL/CODEINE PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE HCL/HYDROCODONE PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE PYRILAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BT PYRILAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE |

# Appendix A Nonbiologics

# Glucocorticoids

| Ingredient code | |
|---------------------------|----------------------|
| P5AR - prednisone | P5BC - dexamethasone |
| P5CB - triamcinolone | P5BB - betamethasone |
| P5AM - methylprednisolone | P5BL - budesonide |
| P5AB - hydrocortisone | P5AH - prednisolone |
| P5AA - cortisone | |